# Randomisierte, multizentrische Studie zum Vergleich der roboterassistierten und der konventionellen laparoskopischen radikalen Prostatektomie

## **LAP-01**

Studienprotokoll Klinische Prüfung nach §23b MPG

Protokoll-Code: LAP-01

Version 3.0

27. Februar 2014

**VERTRAULICHE INFORMATION** 

Das vorliegende Dokument ist vertraulich zu behandeln und darf ohne vorherige schriftliche Genehmigung von Prof. Dr. med. Jens-Uwe Stolzenburg weder vollständig noch in Auszügen an Dritte weitergegeben werden.

## Randomisierte, multizentrische Studie zum Vergleich der roboterassistierten und der konventionellen laparoskopischen radikalen Prostatektomie

Protokoll-Code: LAP-01

Version 3.0

27. Februar 2014

Ich habe das vorliegende Protokoll gelesen und erkläre mich damit einverstanden, die darin enthaltenen Bestimmungen einzuhalten. Ich werde den mir unterstellten Studienmitarbeitern sowie meiner örtlichen Ethikkommission Exemplare dieses Protokolls sowie alle relevanten Informationen zur Verfügung stellen. Ich werde dieses Material mit ihnen besprechen und dafür sorgen, dass sie hinsichtlich der Durchführung der Studie gemäß diesem Protokoll, der lokalen Gesetze und der Deklaration von Helsinki umfassend informiert sind.

| Name des Studienzentrums | |
|-------------------------------|-------|
| Unterschrift des Hauptprüfers | Datum |

## Synopsis

| Titel der Studie | Randomisierte, multizentrische Studie zum Vergleich der roboterassistierten und der konventionellen laparoskopischen radikalen Prostatektomie |
|---|---|
| Kurzbezeichnung der Studie | LAP-01 |
| Indikation | Lokal begrenztes Prostatakarzinom |
| Primäres Ziel der Studie | Kontinenz R-LRPE vs. LRPE Untersuchung, ob bei der Behandlung des lokalen Prostatakarzinoms bis 3 Monate nach einer roboterassistierten laparoskopischen radikalen Prostatektomie (R-LRPE) ein höherer Anteil kontinent ist als nach einer konventionellen laparoskopischen radikalen Prostatektomie (LRPE). Zeit bis zur Erreichung der Kontinenz bis 3 Monate posto- |
| Primärer Endpunkt | perativ |
| Sekundäre Ziele der Studie | Vergleich funktioneller Ergebnisse: R-LRPE vs. LRPE - Kontinenz (ICIQ-SF): 1, 3, 6, 12 Monate p.o Kontinenz (PAD-Verbrauch/Tag): 1, 6, 12 Monate p.o Erektile Funktion (IIEF-5): 3, 6, 12 Monate p.o Residuale Erektile Funktion (REF): 3, 6, 12 Monate p.o. |
| | Vergleich von Lebensqualität, psychosozialem Befinden und Patientenzufriedenheit: R-LRPE vs. LRPE - Gesundheitsbezogene Lebensqualität (EORTC QLQ-C30) 1, 3, 6, 12 Monate p.o Prostataspezifische Lebensqualität (EORTC QLQ-PR25): 3, 6, 12 Monate p.o.; Urinary Symptom Scale: zusätzlich 1 Monat p.o Angst- und Depressivität (HADS): 1, 3, 6, 12 Monate p.o Patientenzufriedenheit: 1, 3, 6, 12 Monate p.o. |
| | Vergleich klinischer Parameter: R-LRPE vs. LRPE - perioperative Parameter: Blutverlust, Transfusionsrate, OP-Zeit (Andockzeit, Prostatektomiezeit, Lymphadenektomiezeit); intraoperative Komplikationen - postoperative Parameter: Residualtumor, postoperative Komplikationen, Krankenhausverweildauer |
| | Vergleich des onkologischen Ergebnisses: R-LRPE vs. LRPE - Rezidivrate mittels PSA-Wert: 3, 6, 12, 24, 36 Monate p.o adjuvante Therapien, diagnostizierter Rezidive, Metastasen (12, 24, 36 Monate p.o.) |
| | Weitere Ziele: - Veränderung von ICIQ, IIEF und Lebensqualität im zeitlichen Verlauf - Einflussfaktoren der Kontinenz |
| Sekundäre Endpunkte | - Kontinenz<br>- Erektile Funktion<br>- Lebensqualität |

### - Angst- und Depressivität - Patientenzufriedenheit - Klinische Parameter - Onkologisches Ergebnis - zweiarmige Studie, kontrolliert, randomisiert, patientensei-Studiendesign tig verblindet, multizentrisch **Arm I** roboterassistierte laparoskopische radikale Prostatektomie (R-LRPE) **Arm II** konventionelle laparoskopische radikale Prostatektomie (LRPE) Randomisierung Arm I: Arm II = 3:1 Visitenzeitpunkte - Baseline (1-2 Tage vor OP) - 1, 3, 6, 12, 24, 36 Monate postoperativ Studienpopulation Einschlusskriterien Histologisch gesichertes Prostatakarzinom (Erstdiagnose) Indikation zur primär-kurativen radikalen Prostatektomie Patientenalter ≤ 75 Jahre (Zeitpunkt der OP) • Patient ist mit Randomisierung einverstanden - Patient ist in der Lage, die Studien-Fragebögen selbständig auszufüllen Durchgeführte und dokumentierte Patientenaufklärung durch einen Prüfarzt Schriftliche Einwilligungserklärung des Patienten zur Teilnahme an der Studie (vor der Randomisierung) Ausschlusskriterien Unzureichende Deutschkenntnisse Schwere kognitive Beeinträchtigungen Adipöse Patienten mit einem BMI > 35 Aktuell vorliegende schwere Begleiterkrankung (z.B. Leberzirrhose, Zweitmalignom bzw. Rezidive jeder Art) Tumorstadium: T4 Früheres Malignom (≤ 3 Jahre vor Einschluss in diese Studie) Neoadjuvante Therapie (Hormontherapie) (≤ 3 Monate vor Einschluss in diese Studie) Patient ist immunkompromittiert (z.B. Organtransplantation, Leukämie) Proband hat eine Vorgeschichte von intermittierender Selbstkatheterisierung (im letzten Jahr vor dem Datum seiner Einwilligungserklärung) Erkrankung an Demenz, chronischer Depression, Psychosen Folgende Behandlungen in den vergangenen 3 Monaten: Operationen am Sigma, ausgedehnte Hämorrhoidalresektion, Transurethrale Nadel Ablation der Prostata (TUNA), Osteosynthese-Versorgungen des Beckenbereiches, Salvage Prostatektomie (Prostatavorbestrahlung),

| | <ul> <li>Patienten mit chronischem Harnwegsinfekt (nachweislich mehr als 5 antibiotikapflichtige Infektionsepisoden im letzten Jahr)</li> <li>Dialysepflichtige Patienten</li> <li>Fehlende Bereitschaft zur Speicherung und Wiedergabe der persönlichen Krankheitsdaten im Rahmen des Protokolls</li> </ul> |
|---|---|
| Patientenzahl | Patienten mit der Indikation im Zeitraum: $N_V$ = 2307<br>Patienten Randomisiert: $N_R$ = 782 Patienten<br>Auswertungspopulation: $N_A$ = 704 Patienten<br>Rando-Verhältnis (R-LRPE) 3 : 1 (LRPE) |
| Therapie | Konventionelle oder roboterassistierte laparoskopische radikale Prostatektomie |
| Messungen | PAD-Verbrauch/Tag, Aktivitätslevel, Trinkmenge; Patienten-<br>fragebögen (ICIQ, IIEF-5, EORTC QLQ-PR25, EORTC<br>QLQ-C30, REF, HADS, Patientenzufriedenheit), PSA, Pros-<br>tatavolumen |
| Biometrie | stratifizierte Randomisation, Deskription der Studienkohorte bzw. der –arme, Time-to-event-Analyse (primärer EP) $\chi^2$ -Test für Proportionen (kategoriale Merkmale) bzw. Rangtests für kontinuierliche Größen (U- bzw. H-Test), ANOVA mit Messwiederholungen für Längsschnittbetrachtungen, allgemeine / verallgemeinerte lineare Modelle |
| Zeitplan | Patientenbezogen - Dauer der Therapie (OP-Zeit): 1 bis 4 Stunden - Nachbeobachtungsdauer: 36 Monate Studienbezogen - Beginn: 2014 - Rekrutierungsdauer: 36 Monate - Gesamterhebungsdauer: 60 Monate - Vorbereitungs-/Auswertungsdauer: 6 Monate |
| Prüfzentren | 4 Zentren (Universitätsklinikum Leipzig, Universitätsklinikum Düsseldorf, Universitätsklinikum Heidelberg, Klinikum Dortmund) |

#### Ablaufdiagramm/Flow Chart



Tabelle 1 Study Schedule

| Ereignis | Screening | | | Behandlun | g und Nachbeok | achtungstermine | • | |
|---|---|---|---|---|---|---|---|---|
| Maßnahme | Prä-OP<br>Baseline | peri-<br>operativ | <b>1 Mo p.o.</b> (30±10 d) follow-up | <b>3 Mo p.o.</b> (90±10 d) follow-up | <b>6 Mo p.o.</b> (180±20 d) follow-up | <b>12 Mo p.o.</b> (365±30 d) follow-up | <b>24 Mo p.o.</b> (730±60 d) follow-up | <b>36 Mo p.o.</b> (1095±60 d) follow-up |
| | Klinik | Klinik | zu Hause | zu Hause | zu Hause | zu Hause | zu Hause | zu Hause |
| CRF Visiten No. | V0 | OP | V1 | V2 | V3 | V4 | V5 | V6 |
| Prüfung PREFERE-Resultat <sup>1</sup> | Х | | | | | | | |
| Einwilligungserklärung nach erfolgter Aufklärung | х | | | | | | | |
| Ein-/ Ausschlusskriterien | Х | | | | | | | |
| Randomisation | Х | | | | | | | |
| Soziodemografie | Х | | | | | | | |
| Anamnese | Х | | | | | | | |
| Karnofsky Performance Status | Х | | | | | | | |
| Begleiterkrankungen | Х | | | | | | | |
| Begleitmedikation <sup>2</sup> | Х | Х | Х | Х | Х | Х | | |
| Verfahrensparameter (perioperative, klinische Daten) | | х | | | | | | |
| PAD-Verbrauch <sup>3</sup> | х | | Х | Х | Х | Х | | |
| ICIQ | Х | | Х | Х | Х | Х | | |
| IIEF-5 | Х | | | Х | Х | Х | | |
| REF | Х | | | Х | Х | Х | | |
| EORTC QLQ-C30 | X | | Х | Х | Х | X | | |
| EORTC QLQ-PR25 | X | | x <sup>7</sup> | Х | Х | Х | | |
| HADS | Х | | Х | Х | Х | Х | | |
| Patientenzufriedenheit | | | Х | X | Х | X | | |
| Aktivitätslevel, Trinkmenge | Х | | Х | Х | Х | Х | | |
| PSA⁴ | Х | | | Х | Х | X | Х | X |
| Kreatinin im Serum <sup>5</sup> | Х | | | | | | | |
| Beurteilung unerwünschter Ereignisse <sup>6</sup> | | x | | | | | | |

Mo = Monate, p.o. = postoperativ ; d = Tage

LAP-01 Version 3.0 / 27.02.2014 Seite 7 von 48

<sup>&</sup>lt;sup>1</sup> Zunächst Aufklärung des Patienten im beteiligten Zentrum für PREFERE-Studie. Patienten, die nicht teilnehmen oder für RPE randomisiert wurden, können für LAP-01 rekrutiert werden.

<sup>&</sup>lt;sup>2</sup> Ab 1 Monat p.o. ausschließlich Informationen über Medikamente, die sich auf die Urogenitalfunktion auswirken sowie potenzsteigernde Hilfsmittel (Viagra, etc.).

<sup>&</sup>lt;sup>3</sup> Tagebuch zu PAD-Verbrauch, Aktivitätslevel und Trinkmenge vom 1. Tag nach Katheterentfernung bis 3 Monat p.o. mit täglicher Eintragung. 6, 12 Monate p.o. einmalige Erfassung des PAD-Verbrauchs. <sup>4</sup> Liegt im Zeitraum von 90 Tagen vor dem Datum der Einwilligungserklärung eine PSA-Datendokumentation vor, kann diese bei der Baseline-Messung berücksichtigt werden. <sup>5</sup> Wird routinemäßig vor OP abgenommen <sup>6</sup> Erfassung unerwünschter Ereignisse während des Klinikaufenthaltes (stationär). <sup>7</sup> Ausschließlich Urinary Symptom Scale.

## Inhaltsverzeichnis

| 1 | Allge | emeine Informationen | 11 |
|---|---|---|---|
| | 1.2 | Protokollidentifizierung<br>Beteiligte Personen und Institutionen<br>Zusammenfassung | 11 |
| 2 | Ratio | onale | 13 |
| | | Forschungsstand und Fragestellung<br>Nutzen-Risiko-Bewertung | |
| 3 | Stud | ienziele | 16 |
| | | Primäres Ziel der Studie/ Primärer EndpunktSekundäre Ziele der Studie/ sekundäre Endpunkte | |
| 4 | Stud | ienbeschreibung | 18 |
| | 4.2<br>4.3<br>4.4 | Studiendesign Personelle und technische Anforderungen Teilnehmende Prüfzentren und Zahl der Patienten Erwartete Studiendauer Studienabbruch Abbruch der Studie in einem Prüfzentrum Abbruch der gesamten Studie bzw. einzelner Studienarme | 18<br>20<br>20 |
| 5 | Stud | ienpopulation | 21 |
| | | Einschlusskriterien<br>Ausschlusskriterien | |
| 6 | Prüf | therapie | 22 |
| 7 | Indiv | ridueller Studienablauf | 23 |
| | 7.2<br>7.3<br>7.3.1<br>7.3.2<br>7.3.3<br>7.3.4<br>7.3.5<br>7.4<br>1<br>7.4.2<br>7.4.3<br>7.4.4<br>7.4.5 | Aufklärung und Einwilligung Aufnahme in die Studie Beschreibung des Studienablaufs Randomisation Datenerhebung zur Baseline Chirurgischer Eingriff und perioperative Datenerhebung Datenerhebung zu den Follow-up-Visiten Vorzeitiger Abbruch der Studientherapie oder der Nachbeobachtung Datenerfassung Kontinenz: PAD-Verbrauch Patienten-Fragebögen Klinische Daten Onkologische Daten Medikamente Vorzeitiger Abbruch für Studienpatienten | 2324252627272729 |
| 8 | | wünschte Ereignisse (AE/SAE/Vorkommnis) | |
| • | 8.1<br>8.1.1<br>8.1.2 | Unerwünschtes Ereignis - AE Definition | 30<br>30<br>30 |

| 8.2<br>8.3 | 2.2 Dokumentations- und Meldeverpflichtungen für den Prüfer Vorkommnis | 31 |
|---|---|---|
| 8.3 | | |
| | 3.2 Meldeverpflichtungen für den Prüfer | |
| 8.4 | Sicherheitsanalysen | |
| 8.5 | Begleiterkrankungen | 32 |
| 8.6 | Therapeutische Maßnahmen | |
| 8.7<br>8.8 | Korrektive Maßnahmen Klassifikation unerwünschter Ereignisse | |
| o.o<br>8.8 | <del>-</del> | |
| 8.8 | | |
| 8.8 | | |
| 8.8 | | |
| 8.8 | 3.5 Ausgang des unerwünschten Ereignisses | 35 |
| 9 Bi | ometrie | 35 |
| 9.1 | Randomisationsalgorithmus | 35 |
| 9.2 | Endpunkte der Studie | 35 |
| _ | 2.1 Primärer Endpunkt | |
| | 2.2 Sekundäre Endpunkte | |
| 9.3<br>9.3 | Statistische Formulierung der Studienfrage | |
| 9.4 | Fallzahldiskussion | |
| 9.4 | | |
| 9.4 | | |
| 9.4 | | |
| 9.4 | | |
| | Verfahren zur Datenanalyse | |
| 9.5<br>9.5 | · | |
| 9.6 | Zwischenauswertungen | |
| 9.7 | Endauswertung | |
| 10 Da | itenmanagement | 39 |
| | _ | |
| 10.1<br>10.2 | Prüfbögen (Case Report Forms - CRF) Datenmanagement | 39 |
| 10.2 | Archivierung | |
| | • | |
| 11 Qւ | ıalitätssicherung | |
| 11.1 | Zugang zu Quelldaten | |
| 11.2 | Monitoring | 41 |
| 12 Et | hische und regulatorische Grundlagen | <b>4</b> 1 |
| 12.1 | GCP-Erklärung | 41 |
| 12.2 | Antragstellung | |
| 13 Ge | esetzliche und administrative Regelungen | 42 |
| 13.1 | Studiendurchführung nach Prüfplan | 42 |
| 13.2 | Nachträgliche Prüfplanänderungen | 42 |
| 13.3 | Verantwortlichkeit der Prüfer und Prüferverträge für klinische Studien | 43 |
| 13.4 | Finanzierung und Versicherungen | |
| 13.5 | Publikationsvereinbarungen und Registrierung | 43 |
| 14 l if | eratur | 45 |

#### Abkürzungsverzeichnis

DGU Deutsche Gesellschaft für Urologie
E-/A-Kriterien Einschluss-/Ausschlusskriterien
EAU European Association of Urology

EERPE Endoskopische extraperitoneale radikale Prostatektomie

EORTC European Organization for Research and Treatment of Cancer

HADS Hospital Anxiety and Depression Scale

ICIQ-SF International Consultation on Incontinence Questionnaire - Short Form

IIEF International Index of Erectile Function

ISF Investigator Site File

LPO Last patient out

LRPE Laparoskopische radikale Prostatektomie

ORPE Offene radikale Prostatektomie

PCA Prostatakarzinom

p.o. Postoperativ

PSA Prostataspezifisches Antigen

QLQ – C30 Quality of Life Questionnaire – Core 30

QLQ – PR25 Quality of Life Questionnaire – Prostate Modul

REF Residuale Erektile Funktion

R-LRPE Roboterassistierte laparoskopische radikale Prostatektomie

RPE Radikale Prostatektomie

## 1 Allgemeine Informationen

## 1.1 Protokollidentifizierung

Protokoll-Code: LAP-01 EudraCT-Nr.: entfällt

Datum der Protokollversion: 27.02.2014

## 1.2 Beteiligte Personen und Institutionen

| STUDIENLEITUNG | |
|---|---|
| Leiter Klinische Prüfung | Prof. Dr. med. Jens-Uwe Stolzenburg FRCS (Ed), FRCS (Eng) Direktor der Klinik und Poliklinik für Urologie Universitätsklinikum Leipzig Liebigstr. 20, 04103 Leipzig Tel: +(49) 341 9717600; Fax. +(49) 341 9717609 Jens-Uwe.Stolzenburg@medizin.uni-leipzig.de |
| Projektmanagement | Dr. phil. Sigrun Holze Studienmanagement, Klinik und Poliklinik für Urologie Universitätsklinikum Leipzig Liebigstr. 20, 04103 Leipzig Tel: +(49) 341 9717629; Fax: +(49) 341 9717609 Mail: Sigrun.Holze@medizin.uni-leipzig.de |
| BIOMETRIE | Dr. rer. nat. Meinhard Mende Biometriker, Zentrum für Klinische Studien Universität Leipzig Härtelstraße 16-18, 04107 Leipzig Tel: +(49) 341 9715770; Fax: +(49) 341 97 16189 Mail: Meinhard.Mende@zks.uni-leipzig.de |
| PRÜFZENTREN | Prof. Dr. med. Jens-Uwe Stolzenburg, FRCS (Ed), FRCS (Eng) Direktor der Klinik und Poliklinik für Urologie Universitätsklinikum Leipzig Liebigstr. 20, 04103 Leipzig Tel: +(49) 341 9717600; Fax. +(49) 341 9717609 Mail: Jens-Uwe.Stolzenburg@medizin.uni-leipzig.de Prof. Dr. med. Markus Hohenfellner Direktor der Klinik für Urologie |
| | Universitätsklinikum Heidelberg<br>Im Neuenheimer Feld 110, 69120 Heidelberg<br>Tel. +(49) 6221 566321; Fax +(49) 6221 565366<br>Mail: Markus.Hohenfellner@med.uni-heidelberg.de |

| | 1 |
|---|---|
| | Prof. Dr. med. Peter Albers Direktor der Klinik für Urologie Universitätsklinikum Düsseldorf Moorenstr. 5, 40225 Düsseldorf Tel. +(49) 211 8118110; Fax: +(49) 211 8118676 Mail: Peter.Albers@med.uni-duesseldorf.de Prof. Dr. med. Michael C. Truß Direktor der Urologischen Klinik Klinikum Dortmund gGmbH Münsterstr. 240, 44145 Dortmund Tel. +(49) 231 95318700; Fax +(49) 231 95318790 Mail: Michael.Truss@klinikumdo.de |
| DATENBANK | André Rothe Zentrum für Klinische Studien Leipzig – KKS Universität Leipzig Härtelstraße 16-18, 04107 Leipzig Tel: +(49) 341 9716 118 Mail: Andre.Rothe@zks.uni-leipzig.de |
| MONITORING | Nicole Köppe-Bauernfeind Zentrum für Klinische Studien Leipzig – KKS Universität Leipzig Härtelstraße 16-18, 04107 Leipzig Tel: +(49) 341 9716 266 Mail: Nicole.Bauernfeind@zks.uni-leipzig.de |
| Gesamtverantwortlicher im<br>Sinne des SPONSORs | Universität Leipzig<br>Ritterstr. 26<br>04109 Leipzig |

#### 1.3 Zusammenfassung

Das Ziel der randomisierten, multizentrischen Studie ist der Vergleich der roboterassistierten laparoskopischen radikalen Prostatektomie (R-LRPE) und der konventionellen laparoskopischen radikalen Prostatektomie (LRPE) hinsichtlich der zentralen Ergebnisparameter. Die R-LRPE hat in den letzten Jahren in zunehmendem Maße Anwendung bei der Behandlung des lokal begrenzten Prostatakarzinoms (PCA) gefunden, wobei ein Vorteil dieser Behandlungsmethode im Vergleich zur LRPE bisher nicht belegt ist, da randomisierte, kontrollierte Vergleichsstudien (RCT) fehlen. Die unsichere Datenlage bezüglich des besten Operationsverfahrens sowohl hinsichtlich des klinischen und onkologischen Behandlungsergebnisses als auch der möglichst schnellen Wiedererlangung der Kontinenz und erektilen Funktion durch den Patienten ist daher ein großes Defizit in der chirurgischen Behandlung des klinisch lokalisierten PCA.

Primärer Endpunkt der Studie ist die Zeit bis zur Wiedererlangung der Kontinenz. Sekundäre Endpunkte sind klinische Parameter und onkologische Tumorkontrolle, erektile Funktion, gesundheitsbezogene und prostataspezifische Lebensqualität, Patientenzufriedenheit sowie psychosoziale Befindlichkeit.

#### 2 Rationale

#### 2.1 Forschungsstand und Fragestellung

Das Prostatakarzinom (PCA) ist der häufigste bösartige Tumor des Mannes. Pro Jahr werden in Deutschland mehr als 60.000 Fälle neu diagnostiziert (RKI 2010). Die Therapie der Wahl beim organbegrenzten Prostatakrebs ist die radikale Prostatektomie (RPE). Die wesentlichen Ziele der RPE sind ein onkologisch gutes Ergebnis mit möglichst wenig positiven Schnitträndern und einer geringen PSA-Rezidivrate sowie ein gutes funktionelles Outcome, d.h. eine möglichst schnelle und vollständige Kontinenz und erfolgreiche Regeneration der erektilen Funktion bei Nerverhalt. Für die Durchführung der RPE stehen verschiedene etablierte Verfahren zur Verfügung. Sie unterscheiden sich in der Operationstechnik und im operativen Zugangsweg (Stolzenburg et al. 2011). Neben den offenen Verfahren haben sich minimal invasive laparoskopische/endoskopische Verfahren durchgesetzt. Die neueste Entwicklung stellt die Kombination aus Laparoskopie und Roboter-System dar.

Das DaVinci Surgical System<sup>TM</sup> der Firma Intuitive Surgical ist das Robotiksystem zur Durchführung von laparoskopischen Eingriffen. Fürsprecher des Systems betonen, dass diese Roboterunterstützte OP-Technik das Armamentarium in der minimal-invasiven Chirurgie mit bisher noch nicht dagewesenen Möglichkeiten hinsichtlich Visualisierung und Präzision erweitert, was zugleich mit besseren Ergebnissen für den Patienten assoziiert wird. Als weiterer Vorteil gilt der höhere ergonomische Komfort für den Operateur, was eine Ermüdung verzögert. Ein Nachteil des DaVinci Systems ist das Fehlen eines taktilen Feedbacks, welches bei der konventionellen Laparoskopie noch teilweise gegeben ist. Zudem ist das System zwar in die meisten OP-Säle integrierbar, jedoch insgesamt relativ groß und unhandlich. Kritiker betonen aber insbesondere die hohen Kosten dieses OP-Verfahrens. Auf Grund der Monopolstellung der Fa. Intuitive Surgical sind die Anschaffungs- und Folgekosten des Da-Vinci Systems gegenüber dem konventionellen Verfahren wesentlich höher.

Unabhängig von diesem Disput hat sich das System in der Urologie fest etabliert. Am häufigsten wird es derzeit bei der RPE zur Therapie des PCA angewendet. In den USA werden mehr als drei Viertel aller radikalen Operationen beim PCA auf diese Weise durchgeführt. Auch in Europa und Deutschland hat das roboterassistierte System in den letzten Jahren eine wachsende Ausbreitung erfahren.

Veröffentlichungen hinsichtlich Tumorkontrolle, postoperativer Kontinenz und Potenz, den Qualitätskriterien der RPE, heben dabei meist positive Ergebnisse des roboterassistierten Verfahrens hervor. Gemäß dem Slogan "besser operiert, schneller gesund und mit besseren Ergebnissen" (Hakenberg 2010) wird für die roboterassistierte Prostatektomie geworben. Dem gegenüber steht die existierende Forschungsrealität. Vergleichsdaten mit der konventionellen Laparoskopie sind rar. Ein Vorteil der roboterassistierten laparoskopischen radikalen Prostatektomie (R-LRPE) im Vergleich zur konventionellen laparoskopischen radikalen Prostatektomie (LRPE) ist bisher nicht belegt, da randomisierte, kontrollierte Vergleichsstudien fehlen. Bei bisher publizierten Berichten handelt es sich vor allem um nichtrandomisierte, unkontrollierte Studien, wobei in den meisten Fällen ein retrospektives Design zugrunde liegt. Darüber hinaus sind Schlussfolgerungen für wichtige Ergebnisparameter wie rezidivfreies Überleben, Kontinenz- und Potenzraten durch kurze Nachbeobachtungszeiten, Unterschiede in den Nachbeobachtungsmethoden und eine fehlende Standardisierung (z.B. hinsichtlich der Messung zentraler Zielkriterien wie Kontinenz) erschwert (S3 Leitlinien, DGU 2011). Der Mangel an randomisierten kontrollierten Studien zum Vergleich der R-LRPE und der LRPE stellt damit ein großes Defizit in der Literatur zur chirurgischen Behandlung des lokalisierten PCA dar.

Wie ein systematisches Review in der Zeitschrift European Urology belegt, ist die publizierte Literatur vor allem auf Beobachtungsstudien von zum Teil geringer wissenschaftlicher Qualität begrenzt (Kang et al. 2010). Von insgesamt 75 begutachteten Originalarbeiten waren 75% Fallstudien, 11 (15%) retrospektive Studien und nur zwei (2,7%) randomisierte, kontrollierte Studien. Die beiden randomisierten Untersuchungen konzentrierten sich dabei nicht auf den Vergleich der R-LRPE zur LRPE oder zur offenen RPE, sondern auf technische Modifikationen der R-LRPE. Deutlich wurde bei der Analyse zudem, dass allein 12 Autoren an 72% (54 von 75) der veröffentlichten Artikel beteiligt waren.

Asimakopoulos et al. (2011) vergleichen in der ersten randomisierten, monozentrischen Studie mit insgesamt nur 64 Patienten pro Untersuchungsgruppe (LRPE vs. R-LRPE) die klinischen, funktionellen und onkologischen Ergebnisse beider Methoden. Bezüglich der perioperativen Daten (Operationszeit, Blutverlust) und der Komplikationen gibt es keine signifikanten Unterschiede. Auch die Kontinenzrate nach 3, 6 und 12 Monaten unterscheidet sich nicht signifikant zwischen beiden Gruppen (LRPE: 63%, 75% 83% vs. R-LRPE: 69%, 88%, 94%). Während sich 3 und 6 Monate postoperativ keine signifikanten Unterschiede in der erektilen Funktion finden, zeigt die R-LRPE 12 Monate postoperativ bessere Ergebnisse (32% bei LRPE vs. 77 % bei R-LRPE, P < 0.0001). Für eine randomisierte Studie zum Vergleich beider Methoden ist eine Patientenzahl von 64 Patienten pro Methode allerdings gering. Anzumerken bleibt außerdem, dass die Potenzrate der LRPE-Gruppe mit 32% niedrig im Vergleich zu bisher publizierten LRPE-Daten ist (Rassweiler et al. 2006; Badani et al. 2007; Krambeck et al. 2009; Murphy et al. 2009; Patel et al. 2010). Die Potenzrate der R-LRPE-Gruppe ist so hoch wie publizierte Daten zur LRPE (ebd.).

Auch Ficarra et al. (2009) kommen in ihrem systematischen Review mit kumulativer Analyse zu dem Schluss, dass sich anhand vorhandener Daten kein Beleg für den Vorteil eines der Operationsverfahren (LRPE vs. R-LRPE) bzgl. funktioneller und onkologischer Ergebnisse ergibt. Sie verweisen deutlich auf das Fehlen randomisierter Studien. Resümierend betonen die Autoren, dass es aufgrund der vorliegenden Datenbasis dringend prospektiver, multizentrischer Studien bedarf, um die Wertigkeit neuer urologischer OP-Methoden im Vergleich zu etablierten Verfahren evident messen zu können.

Unser Studienprotokoll zielt darauf ab, die bestehende Forschungslücke zu schließen. Ob die R-LRPE im Vergleich zur konventionellen Laparoskopie tatsächlich zu einer Verbesserung der Ergebnisse bei der RPE führt, kann nur durch eine klinische Studie geprüft werden, wie sie mit dem vorliegenden Antrag geplant ist. Das Ziel unserer randomisierten, kontrollierten, multizentrischen Studie ist daher ein umfassender Vergleich der R-LRPE und der LRPE. Primärer Endpunkt ist die Zeit bis zur Wiedererlangung der Kontinenz. Sekundäre Endpunkte sind klinische Parameter und onkologische Tumorkontrolle, erektile Funktion, gesundheitsbezogene und prostataspezifische Lebensqualität, Patientenzufriedenheit sowie psycho-

soziale Befindlichkeit (Angst und Depressivität).

In den vier beteiligten Prüfzentren (Universitätsklinikum Leipzig, Universitätsklinikum Heidelberg, Universitätsklinikum Düsseldorf, Klinikum Dortmund) werden zusammen jährlich annähernd 1000 Patienten prostatektomiert. Zudem werden in diesen Kliniken sowohl die LRPE als auch die R-LRPE angewandt, was eine Randomisierung ermöglicht. Darüber hinaus kann auf die Erfahrungen verschiedener prospektiver Studien zurückgriffen werden. So arbeiteten wir unter anderem an einer Vergleichsstudie zur Lebensqualität nach radikaler Prostatektomie, die zwischen 2007 und 2010 von der Deutschen Krebshilfe gefördert wurde. Im Rahmen dieser prospektiven, multizentrischen Studie wurden Patienten aus sieben Kliniken einbezogen. Ziel war der Vergleich zwischen laparoskopischer/endoskopischer radikaler Prostatektomie und offener radikaler Prostatektomie bezüglich funktioneller und lebensqualitätsbezogener Daten (Holze et al. 2011, Köhler. et al. 2011). Das aktuelle Studienvorhaben greift das bewährte validierte Instrumentarium dieser Studie auf und erweitert es.

Zusammengefasst vereinigt unser Forschungsvorhaben folgende Vorteile:

- Erste randomisierte, multizentrische Studie weltweit, die R-LRPE und LRPE vergleicht
- Umfassende prä-, peri- und postoperative Evaluierung klinischer, onkologischer, funktioneller, lebensqualitätsbezogener und psychosozialer Daten
- Evaluierung anhand validierter Messinstrumente
- Beurteilung verschiedener Verfahren zur Messung von Kontinenz (PAD-Tagebuch, ICIQ-SF, EORTC QLQ-PR25 Urinary Symptom Scale)

Die Studie soll wesentlich zu einer validen Datenbasis des roboterassistierten Operationsverfahrens in der Urologie beitragen. Aus dem Blickwinkel des Nutzen-Risiko-Kosten Verhältnisses ist zu fragen, ob sich der finanzielle Mehraufwand durch den DaVinci® Roboter auch in einem besseren Outcome wiederspiegelt. Die Studienergebnisse zielen auf eine objektive und kritische Beantwortung der Frage, ob die R-LRPE im Vergleich zu konventionellen laparoskopischen Methode tatsächlich einen Vorteil in der Behandlung des lokalen Prostatakarzinoms einnimmt. Valide Vergleichsdaten der beiden operativen Verfahren sind unerlässlich für evidenzbasierte Therapieentscheidungen.

#### 2.2 Nutzen-Risiko-Bewertung

Sowohl die LRPE als auch die R-LRPE sind zur Behandlung des lokal begrenzten Prostatakarzinoms sicher und wirksam. Ihre klinische Wirksamkeit und Sicherheit sind in der Fachliteratur hinreichend belegt (S3 Leitlinie der DGU 2011). Bei beiden OP-Methoden handelt es sich um Standardbehandlungen in der Urologie. Die R-LRPE führt im Vergleich zur LRPE zu keiner Zusatzbelastung für den Patienten. Der DaVinci® Roboter ist ein zugelassenes Medizinprodukt, das in der geplanten Indikation ohne zusätzliche, studienbedingte invasive Maßnahmen verwendet wird. Da es die Hypothese ist, dass es den Patienten nach einer R-LRPE schneller besser geht, erhält der Patient durch das gewählte Randomisationsverhältnis (3 : 1 = R-LRPE : LRPE) eine größere Chance, roboterassistiert operiert zu werden (vgl. Randomisation, Kapitel 7.3.1).

Die 3D-Sicht ist zurzeit noch ein Vorteil der roboterassistierten Methode. Inwieweit sich die subjektiv als sehr positiv empfundene 3D-Sicht tatsächlich auf die OP-Technik und damit auch auf die funktionellen Ergebnisse auswirkt, ist allerdings bisher in keiner Weise nachgewiesen. Ein deutlicher Vorteil der R-LRPE im Vergleich zur LRPE ist die geringere Belastung für den Operateur. Dieser sitzt ergonomisch an einer vom Operationstisch distanten Konsole und steuert durch manuelle Bewegung beider Hände die Instrumente. Die ergonomische Sitzhaltung ermöglicht dem Operateur dabei eine entspannte und konzentrierte Operation.

Als Nachteil des DaVinci® Systems gilt das Fehlen eines taktilen Feedbacks. Dieses ist bei der konventionellen Laparoskopie noch partiell vorhanden. Zudem ist das System zwar in die

meisten OP-Säle integrierbar, jedoch insgesamt relativ groß und unhandlich. Kritiker heben insbesondere die hohen Kosten des roboterassistierten OP-Verfahrens hervor. Die Anschaffungs-, Material- und Wartungskosten des DaVinci® Systems sind gegenüber dem konventionellen laparoskopischen Verfahren wesentlich höher. Für die Kliniken entstehen durch die roboterassistierte OP-Methode einerseits Mehrkosten pro Fall (welche bei steigenden Fallzahlen begrenzt werden können), andererseits erfolgt ein Imagegewinn für die Klinik ("schonende Operationsverfahren", "neueste Technologie") (Hakenberg 2010).

Mögliche Risiken beider OP-Methoden (LRPE, R-LRPE) sind u.a. Bildung von Blutgerinnseln (Thrombose, Embolie), Verletzung größerer Blutgefäße / Blutungen, Wundinfektion, Harninkontinenz, erektile Dysfunktion, Infertilität, Anastomoseninsuffizienz, Lymphozele, Nervenreizung / Nervenverletzung, Verletzung des Enddarms, Verletzung / Einengung der Harnleiter, Anastomosenstriktur, Blasenhalsobstruktion, Urethrastriktur, Verbleiben von Tumorgewebe (sog. R1-Resektion, positiver Schnittrand) (S3 Leitlinie der DGU 2011).

Sowohl die LRPE als auch die R-LRPE als minimal invasive Verfahren haben ein geringeres Akzesstrauma und verursachen dadurch geringere systemische Reaktionen als die offene OP. Der intraoperative Blutverlust und die Transfusionsrate sind beim konventionellen und roboterassistierten laparoskopischen Vorgehen geringer (ebd.). Bezüglich des postoperativen biochemischen PSA-Verhaltens zeigen sich im Vergleich der Literatur keine signifikanten Unterschiede zwischen LRPE und R-LRPE (Do et al. 2012).

Diese Studie kommt der medizinischen Gemeinschaft sowie den Patienten zugute, da sie die verhältnismäßige Wirksamkeit für die beiden häufig angewandten chirurgischen Behandlungsmethoden des lokal begrenzten Prostatakarzinoms untersucht. Diese Daten helfen Ärzten wie Patienten, in Zukunft informierte Entscheidungen in Bezug auf die Wahl der PCA-Behandlung zu treffen.

#### 3 Studienziele

Im Rahmen der Studie werden funktionelle, klinische, onkologische und lebensqualitätsbezogene Parameter der roboterassistierten und der konventionellen laparoskopischen radikalen Prostatektomie verglichen.

#### 3.1 Primäres Ziel der Studie/ Primärer Endpunkt

Primäres Ziel der Studie ist es zu untersuchen, ob Patienten nach einer R-LRPE schneller kontinent sind als nach einer LRPE.

Primärer Endpunkt ist die Zeit bis zum Erreichen der Kontinenz bis 3 Monate postoperativ. Dazu wird der tägliche Bedarf an PADs erfasst. Ein Patient gilt dann als kontinent, wenn er an drei aufeinanderfolgenden Zeitpunkten keine PADs mehr benötigt hat. Als Kontrollvariablen werden ebenfalls das Aktivitätslevel und die Trinkmenge des Patienten erhoben.

Gründe für die Wahl des primären Endpunktes:

Der Kontinenzstatus stellt einen zentralen Qualitätsindikator einer radikalen Prostatektomie dar; er misst damit den Erfolg der Operation. Der Erhalt der Harnkontinenz wird auch in den S3-Leitlinie der Deutschen Gesellschaft für Urologie (Punkt 5.15) als Ziel der Prostatektomie angeführt. Das geführte Tagebuch hat dabei entscheidende Vorteile. Niemand kann die Auswirkung der Therapie auf die Kontinenz besser einschätzen als der Patient selbst. Von besonderer Aussagekraft sind Daten, die Rückschlüsse auf den kontinuierlichen Verlauf zulassen. Deshalb sind engmaschige Verlaufsdaten in Form von Eintragungen in das Tagebuch essentiell. Die regelmäßigen Eintragungen ins Patiententagebuch funktionieren dabei wie ein Protokoll.

Die Realisierbarkeit der Kontinenzmessung anhand des PAD-Verbrauchs ist sowohl prä- als auch postoperativ bei allen Patienten gegeben. Die Messung ist nicht invasiv und stellt damit für den Patienten keine zusätzliche Belastung dar. Die tägliche Messung gewährleistet die Abbildung des Verlaufs und berücksichtigt die Realisierung der Messung beim Patienten.

Schaut man sich die Literatur zur Kontinenz nach RPE beider OP-Verfahren an, kommt es nach einer längeren Zeit (> 6 Monate p.o.) meist zu einer Nivellierung der Kontinenzergebnisse (Ficarra et al. 2009). Um einen möglichen Unterschied zwischen den Verfahren auch sehen zu können, ist die frühe postoperative Phase entscheidend, weshalb der Verlauf während der ersten 3-Monate nach dem operativen Eingriff als primärer Endpunkt gewählt wird. Gerade aus Patientensicht ist eine frühe Erreichung der Kontinenz essentiell, da dies einen beträchtlichen Gewinn an Lebensqualität bedeutet. Dies hat deutliche Auswirkungen auf die Gestaltung des Lebensalltags und die (altersabhängige) Möglichkeit einer Rückkehr ins Arbeitsleben. Der harte Endpunkt (Kontinenz = 0 PADs) ermöglicht zudem den Vergleich mit anderen Messmethoden in der Literatur.

- Ethisch: Nicht invasiv, keine Zusatzbelastung für den Patienten
- Klinisch: Unterschiede in der Kontinenz machen für den Patienten einen wesentlichen Unterschied, der Zeitpunkt der Erreichung von Kontinenz ist essentiell für den Patienten
- Biometrisch: Verlässlich messbar, objektiv und reproduzierbar; vergleichbar mit anderen Skalen (z. B. ICIQ-SF = 0); sowohl eine mittlere Zeit bis zum Erreichen von Kontinenz als auch die Raten in beiden Gruppen zu bestimmten Zeitpunkten sind schätzbar
- Logistisch: Lückenlos und mit geringem finanziellen Aufwand bei allen Patienten messbar.

#### 3.2 Sekundäre Ziele der Studie/ sekundäre Endpunkte

Vergleich der funktionellen Ergebnisse: R-LRPE vs. LRPE

- Kontinenz (ICIQ-SF): 1, 3, 6, 12 Monate p.o.
- Kontinenz (PAD-Verbrauch/Tag): 1, 6, 12 Monate p.o.
- Erektile Funktion (IIEF-5): 3, 6, 12 Monate p.o.
- Residuale Erektile Funktion (REF): 3, 6, 12 Monate p.o.

Vergleich von Lebensqualität, psychosozialem Befinden und Patientenzufriedenheit: R-LRPE vs. LRPE

- Gesundheitsbezogene Lebensqualität (EORTC QLQ-C30): 1, 3, 6, 12 Monate p.o.
- Prostataspezifische Lebensqualität (EORTC QLQ-PR25): 3, 6, 12 Monate p.o.; Urinary Symptom Scale: zusätzlich 1 Monat p.o.
- Angst- und Depressivität (HADS): 1, 3, 6, 12 Monate p.o.
- Patientenzufriedenheit: 1, 3, 6, 12 Monate p.o.

#### Vergleich klinischer Parameter: R-LRPE vs. LRPE

- perioperative Parameter: Blutverlust, Transfusionsrate, OP-Zeit (Andockzeit, Prostatektomiezeit, Lymphadenektomiezeit); intraoperative Komplikationen
- postoperative Parameter: R-Klassifikation (Pathologiebefund), postoperative Komplikationen

Vergleich des onkologischen Ergebnisses: R-LRPE vs. LRPE

- Rezidivrate mittels PSA-Wert: 3, 6, 12, 24, 36 Monate p.o.
- Adjuvante Therapien, diagnostizierter Rezidive, Metastasen

#### Weitere Ziele:

- Veränderung von ICIQ, IIEF und Lebensqualität im zeitlichen Verlauf
- potenzielle Einflussfaktoren der Kontinenz

## 4 Studienbeschreibung

#### 4.1 Studiendesign

Es handelt es sich um eine randomisierte, patientenseitig verblindete, multizentrische, zweiarmige klinische Studie nach §23b Medizinproduktegesetz.

Der primäre Endpunkt wird nach drei Monaten erhoben und die Patientennachbeobachtung wird über drei Jahre vorgenommen, um onkologisch relevante Langzeitdaten zu erheben. Die Verblindung wird bis 3 Monate postoperativ aufrechterhalten, danach erfolgt die Entblindung.

#### **Therapiearme**

- Arm I roboterassistierte laparoskopische radikale Prostatektomie (R-LRPE)
- Arm II konventionelle laparoskopische radikale Prostatektomie (LRPE)

#### Randomisierung

Arm I : Arm II = 3 : 1

#### 4.2 Personelle und technische Anforderungen

Bedingungen für die Teilnahme der Prüfzentren an der Studie sind:

- Die Prüfarzte müssen Erfahrung in der Behandlung von Prostatakarzinom-Patienten haben und in der Durchführung von LRPE und/oder R-LRPE die entsprechende Erfahrung aufweisen.
- In Anlehnung an die S3-Leitlinie der Deutschen Gesellschaft für Urologie (2011) soll die radikale Prostatektomie nur unter Leitung eines erfahrenen Operateurs durchgeführt werden. Dies beinhaltet die Durchführung von mindestens 50 Prostatektomien in einer Einrichtung pro Jahr sowie mindestens 25 pro Operateur pro Jahr sowie ein entsprechendes Ausbildungsprogramm.
- Das Studienzentrum verfügt über das geeignete Personal und die angemessene Ausstattung, um das Protokoll durchzuführen und dessen Einhaltung sicherzustellen.
- Die Prüfarzte und das weitere Studienpersonal verpflichten sich, alle geltenden Vorschriften hinsichtlich der Durchführung von klinischen Studien (z. B. Vorschriften der Ethikkommission) zu erfüllen.
- Im Verlauf der Studie werden on-site-Monitoring-Besuche zur Source Data Verification durchgeführt. Hierfür werden die Originaldaten (Krankenakte, Laborblätter, etc.) für eine Überprüfung der Einträge auf den CRFs zur Verfügung gestellt sowie der Zugang zu den Räumlichkeiten der Studiendurchführung ermöglicht.

#### 4.3 Teilnehmende Prüfzentren und Zahl der Patienten

In 2010 und 2011 konnten an den vier teilnehmenden urologischen Kliniken die in Tabelle 2 dargestellten Patientenzahlen (radikale Prostatektomie) erreicht werden. Angesichts steigender Diagnoseraten beim Prostatakarzinom können diese Zahlen auch für den Durchführungszeitraum der Studie angenommen werden. Abzüglich relevanter Ausschlusskriterien wie ungenügende Deutschkenntnisse bzw. Alter ≥75 Jahre sind etwa 80% der Patienten für die Studie geeignet.

#### Universitätsklinikum Leipzig

Prof. Dr. med. Jens-Uwe Stolzenburg Direktor der Klinik und Poliklinik für Urologie

Liebigstr. 20, 04103 Leipzig

#### Universitätsklinikum Heidelberg

Prof. Dr. med. Markus Hohenfellner Direktor der Klinik für Urologie Im Neuenheimer Feld 110, 69120 Heidelberg

#### Universitätsklinikum Düsseldorf

Prof. Dr. med. Peter Albers Direktor der Klinik für Urologie Moorenstr. 5, 40225 Düsseldorf

#### Klinikum Dortmund gGmbH

Prof. Dr. med. Michael C. Truß Direktor der Urologischen Klinik Münsterstr. 240, 44145 Dortmund

Tabelle 2 Anzahl Patienten für laparoskopische radikale Prostatektomie

| | Leipzig | Heidelberg | Düsseldorf | Dortmund | Gesamt |
|---|---|---|---|---|---|
| Anzahl der Patienten in den letzten 2 Jahren 1) | 794 | 330 | 200 | 600 | 1924 |
| Potentielle Patienten pro Jahr 2) | 317 | 132 | 80 | 240 | 769 |

Anzahl der Patienten mit einem lokal begrenzten Prostatakarzinom, die an dem jeweiligen Zentrum in den letzten zwei Jahren eine laparoskopische radikale Prostatektomie erhalten haben

Somit werden jährlich 769 Patienten erwartet, welche die E-/A-Kriterien erfüllen. Die zeitgleich geplante PREFERE-Studie überschneidet sich hinsichtlich des Patientenklientels in Teilen mit der LAP-01-Studie. Daher wird für LAP-01 ein sogenanntes zweistufiges Rekrutierungsmodell festgelegt. Dies bedeutet, dass Patienten unter Berücksichtigung der entsprechenden E-/A-Kriterien zunächst auf ihre Teilnahme an der PREFERE-Studie befragt und randomisiert werden. Erst im Anschluss werden sie ggfs. für die LAP-01 Studie aufgeklärt. Dieses Vorgehen lässt sich wie folgt im Abbildung 1 darstellen:

Abbildung 1: Rekrutierungsschema



Anzahl der Patienten, die in dem jeweiligen Zentrum voraussichtlich pro Jahr für die zur Förderung beantragten Studie rekrutiert werden können; geschätzte 20% erfüllen nicht die E-/A-Kriterien

Patienten, welche die Einschlusskriterien für LAP-01, nicht aber für PREFERE erfüllen sowie Patienten, die eine Studienteilnahme bei PREFERE ablehnen, stellen potentielle Studienpatienten für LAP-01 dar. Zudem stehen die rund 1/4 Patienten, welche in PREFERE für den radikalen Prostatektomie-Arm randomisiert werden, für LAP-01 zur Verfügung (s. Abb. 1).

Nimmt man an, dass durch dieses Vorgehen vom Gesamtaufkommen der vier Kliniken rund 40% der Patienten an der Studie teilnehmen, wären dies ca. 300 pro Jahr. Da die Studienteilnahme für die Patienten kaum einen erhöhten Aufwand bedeutet, wird mit je maximal 10% Drop-Outs bis 3 Monate nach OP bzw. bis zu 12 Monaten nach OP gerechnet.

#### 4.4 Erwartete Studiendauer

Die einzelnen Patienten werden nach Wahrnehmung der letzten Visite (36 Monate postoperativ bzw. 24 Monate postoperativ, vgl. 9.7) aus der Studie entlassen. Vom Aufnahmezeitpunkt des ersten Patienten bis zur letzten Visite des letzten Patienten wird eine Gesamterhebungszeit von 60 Monaten kalkuliert. Die Rekrutierungszeit beträgt 36 Monate.

Für Vorbereitung, Datenauswertung und Berichterstellung werden 6 Monate außerhalb der Erhebungszeit eingeplant. Endauswertung und Publikation der Follow-up Erhebungen bis 12 Monate postoperativ erfolgen im Anschluss an die 12 Monats-Visite des letzten Patienten. Die onkologischen Ergebnisse 24 und 36 Monate postoperativ werden nach der letzten Visite (36 Monate p.o.) des letzten Patienten ausgewertet.

#### 4.5 Studienabbruch

Das Vorgehen beim Abbruch der Studie für einen einzelnen Patienten wird im Kapitel 7.3.5 erläutert.

#### 4.5.1 Abbruch der Studie in einem Prüfzentrum

Die Studie kann in einem Prüfzentrum abgebrochen werden, wenn:

- die Studiendurchführung nicht dem Prüfplan genügt,
- · die Datenqualität unzureichend ist,
- es unzureichend rekrutiert.

Über den Ausschluss entscheidet die Studienleitung, gegebenenfalls in Abstimmung mit dem Biometriker.

Prüfzentren, die nicht mehr an der Studie teilnehmen wollen/können, müssen die Studienleitung unverzüglich über ihre Entscheidung informieren. Die Entscheidung sollte immer begründet werden. Die Weiterbehandlung noch in der Studie befindlicher Patienten wird mit der Studienleitung abgesprochen.

#### 4.5.2 Abbruch der gesamten Studie bzw. einzelner Studienarme

Die Studie kann durch die Studienleitung vorzeitig abgebrochen werden im Falle von:

- schwerwiegenden unerwünschten Ereignissen
- Änderungen in der Nutzen-Risiko-Bewertung, z.B. aufgrund von unerwarteten unerwünschten Ereignissen

- neuen Erkenntnissen aus anderen Studien
- nicht ausreichender Rekrutierungsrate.

Die endgültige Entscheidung über den Abbruch der Studie liegt bei der Studienleitung, ggfs. nach Absprache mit der Biometrie.

## 5 Studienpopulation

In die Studie werden Männer mit Prostatakarzinom entsprechend der Einschlusskriterien aufgenommen. Die Prüfärzte jedes Zentrums müssen prüfen und bestätigen, dass die Patienten alle Einschlusskriterien und keine der Ausschlusskriterien für die Aufnahme in die Studie erfüllen. Die Prüfung der Einschluss- und Ausschlusskriterien muss vor der Randomisierung und dem chirurgischen Eingriff sowie nach der Prüfung des PREFERE-Studien Resultats (s. Flow Chart S. 6; Abbildung 1, S. 19) erfolgen.

#### 5.1 Einschlusskriterien

- Histologisch gesichertes Prostatakarzinom (Erstdiagnose)
- Indikation zur primär-kurativen radikalen Prostatektomie
- Patientenalter ≤ 75 Jahre (Zeitpunkt der OP)
- Patient ist mit Randomisierung einverstanden
- Patient ist in der Lage, die Studien-Fragebögen selbständig auszufüllen
- Durchgeführte und dokumentierte Patientenaufklärung durch einen Prüfarzt
- Schriftliche Einwilligungserklärung des Patienten zur Teilnahme an der Studie (vor der Randomisierung)

#### 5.2 Ausschlusskriterien

- Unzureichende Deutschkenntnisse
- Schwere kognitive Beeinträchtigungen
- Adipöse Patienten mit einem BMI > 35
- Aktuell vorliegende schwere Begleiterkrankung (z.B. Leberzirrhose, Zweitmalignom bzw. Rezidive jeder Art)
- Tumorstadium: T4
- Früheres Malignom (≤ 3 Jahre vor Einschluss in diese Studie)
- Neoadjuvante Therapie (Hormontherapie) (≤ 3 Monate vor Einschluss in diese Studie)
- Patient ist immunkompromittiert (z.B. Organtransplantation, Leukämie)
- Proband hat eine Vorgeschichte von intermittierender Selbstkatheterisierung (im letzten Jahr vor dem Datum seiner Einwilligungserklärung)
- Erkrankung an Demenz, chronischer Depression, Psychosen
- Folgende Behandlungen in den vergangenen 3 Monaten: Operationen am Sigma, ausgedehnte Hämorrhoidalresektion, Transurethrale Nadel Ablation der Prostata (TUNA), Osteosynthese-Versorgungen des Beckenbereiches, Salvage Prostatektomie (Prostatavorbestrahlung).
- Patienten mit chronischem Harnwegsinfekt (nachweislich mehr als 5 antibiotikapflichtige Infektionsepisoden im letzten Jahr)
- Dialysepflichtige Patienten
- Fehlende Bereitschaft zur Speicherung und Wiedergabe der persönlichen Krankheitsdaten im Rahmen des Protokolls

## 6 Prüftherapie

Für die Durchführung der radikalen Prostatektomie (RPE) stehen verschiedene etablierte OP-Verfahren zur Verfügung. Sie unterscheiden sich in der Operationstechnik und im operativen Zugangsweg (Kirby et al. 2007). Aus tumorchirurgischer Sicht sind alle Verfahren als gleichwertig einzustufen (Ficarra et al. 2009).

Das Ziel der RPE ist die vollständige Entfernung der krebsbefallenen Vorsteherdrüse. Hierbei wird die Prostata, die zwischen Harnröhre und Blase liegt, samt Samenblasen und Anteilen der Samenleiter entfernt. Anschließend wird die Blase mit dem Harnröhrenstumpf wieder vernäht. Dieses Prinzip ist bei der konventionellen und der roboter-assistierten laparoskopischen Prostatektomie gleich. Abhängig vom Befund werden in einigen Fällen die Lymphknoten im kleinen Becken ebenfalls entfernt. Des Weiteren kann bei beiden Verfahren der einoder beidseitige Erhalt des neben der Prostata verlaufenden Gefäß-Nerven-Bündels (in Abhängigkeit von der Ausbreitung des Tumors) erfolgen.

Im Unterschied zur offenen retropubischen Prostatektomie werden bei den minimal invasiven laparoskopischen Verfahren lange, dünne chirurgische Instrumente sowie eine Stabkamera für die gesamte Operation verwendet. Das Kamerabild wird vergrößert auf einem Monitor abgebildet (Guillonneau & Vallancien 2000, Stolzenburg et al. 2011). Die laparoskopische Prostatektomie kann transperitoneal oder extraperitoneal erfolgen. In Rückenlagerung und Intubationsnarkose werden halbkreisförmig fünf Trokare in den Unterbauch eingebracht: ein subumbilikaler Zugang für den Kameratrokar und jeweils zwei im Unterbauch befindliche Trokare für die Arbeitsinstrumente.

Die Kombination aus Laparoskopie und Roboter-System (DaVinci®) stellt die neueste Entwicklung dar. Technisch handelt es sich bei dem roboterassistierten System um einen Telemanipulator, d.h. das System führt keine eigenständigen Bewegungen im Patienten durch, sondern folgt lediglich der Handbewegung des Operateurs. Es besteht aus drei wesentlichen Komponenten: der Steuerkonsole, drei oder vier interaktiven, von der Konsole gesteuerten Roboter-Armen und einem Endoskopiesystem. Der Operateur sitzt ergonomisch an einer vom Operationstisch distanten Konsole mit einem 3-dimensionalen High definition-Videosichtsystem. Er steuert durch manuelle Bewegung beider Hände die durch eine ausgefeilte Mikromechanik unterstützten Roboterarme (7 Freiheitsgrade der Instrumente, skalierte Bewegungen, Tremorfilter), welche über rasch austauschbare Mikroinstrumente durch kleine, 8 mm große Trokare in den Bauchraum bzw. extra- und retroperitonealen Raum des Patienten eingeführt werden. Durch einen weiteren Port wird eine 3-dimensionale endoskopische computergesteuerte HD-Videokamera eingeführt, welche das auf dem Monitor wiedergegebene 3D-Bild 10-15fach vergrößert (Guillonneau & Vallancien 2000, Stolzenburg et al. 2011).

Morbidität und Mortalität sind nach der EAU-Leitlinie (Heidenreich et al. 2007) für die radikale Prostatektomie wie folgt angegeben: Therapierelevante Blutung (= major bleeding, 1.0 - 11.5%), Rektale Verletzung (0 - 5,4%), Tiele Beinvenenthrombose (0 - 8,3%), Lungenembolie (0,8 - 7,7%), Lymphozele (0 - 3,0%), Urin-Leckage, Fistel (0,3 - 15,4%), geringradige Belastungsinkontinenz (4,0 - 50,0%), Hochgradige Belastungsinkontinenz (0 - 15,4%), Erektile Dysfunktion (29,0 - 100%), Blasenhalsobstruktion (0,5 - 14,6%), Ureterobstruktion (0 - 0,7), Urethrastriktur (2,0 - 9,0%), peri-operativer Tod (0 - 2.1). Eine detaillierte Dokumentation evaluierter Komplikationen nach LRPE und R-LRPE findet sich auch bei Agarwal et al. (2011) und Hakimi et al. (2011).

Die konventionelle und die roboterassistierte laparoskopische radikale Prostatatektomie sind etablierte Operationsverfahren, die im Rahmen der Studie entsprechend den Operationsstandards in den Prüfzentren durchgeführt werden. Zusätzliche Interventionen außerhalb der routinemäßigen Behandlung erfolgen nicht.

#### 7 Individueller Studienablauf

#### 7.1 Aufklärung und Einwilligung

Die Aufklärung jedes Patienten erfolgt durch ein Gespräch zwischen dem Prüfarzt und dem Patienten vor Einschluss in die Studie. Hierbei wird der Patient über Wesen, erwartete Vorteile und mögliche Risiken informiert. Patienten müssen über ihr Recht aufgeklärt werden, jederzeit aus der Studie ausscheiden zu können, ohne dass ihnen dadurch Nachteile entstehen bzw. Leistungen entgehen, auf die sie ansonsten ein Anrecht haben. Sie müssen außerdem darüber informiert werden, dass ein Ausscheiden aus der Studie ihre zukünftige medizinische Versorgung nicht gefährdet. Der Prüfarzt hat dem Patienten ausreichend Bedenkzeit und Gelegenheit für Rückfragen einzuräumen und muss sich davon überzeugen, dass die Aufklärung vom Patienten verstanden wurde. Alle Fragen des Patienten müssen beantwortet und eventuelle Unklarheiten beseitigt werden. Die Einwilligung des Patienten muss sich ausdrücklich auch auf die Erhebung und Verarbeitung von personenbezogenen Daten beziehen. Deshalb werden die Patienten explizit über Zweck und Umfang der Erhebung und die Verwendung dieser Daten informiert. Der Patient stimmt schriftlich der Speicherung von vollständigen Namen, Geburtsdaten, Adressen, Telefonnummern in der Studienzentrale (Klinik für Urologie, Universitätsklinikum Leipzig) zur späteren Kontaktaufnahme zu. Er stimmt zu, dass seine Daten nach Beendigung oder Abbruch der Studie mindestens zehn Jahre aufbewahrt werden.

Es ist darauf zu achten, dass die Patienten die Einwilligung zur Teilnahme an der Studie selbstständig unterschreiben und datieren. Ein Exemplar der Patientenaufklärung und der unterschriebenen Patienteneinwilligung wird dem Patienten ausgehändigt. Ein weiteres Exemplar verbleibt im Prüfzentrum und wird dort im Studienordner aufbewahrt.

Die Patientenaufklärung und -einwilligung ist im Prüferordner zu finden.

#### 7.2 Aufnahme in die Studie

Patienten mit einer neudiagnostizierten Prostatakrebserkrankung, die in einem der Prüfzentren (Universitätsklinikum Leipzig, Universitätsklinikum Heidelberg, Klinikum Dortmund, Universitätsklinikum Düsseldorf) behandelt werden, die Einschlusskriterien erfüllen und keine Ausschlusskriterien aufweisen, werden nach Aufklärung und Erteilen der Einwilligung konsekutiv in die Studie einbezogen und randomisiert. Alle Studienteilnehmer werden der Studienzentrale (Klinik und Poliklinik für Urologie, Universitätsklinikum Leipzig) gemeldet. Nach jedem eingeschlossenen Studienpatienten erfolgt von den Prüfzentren per Fax (0341 – 97 17679) eine Meldung an die Studienzentrale entsprechend des Registrierungsbogens. Ein Muster des Registrierungsbogens wird in den Prüferordner aufgenommen. Die Rekrutierung der Patienten erfolgt in Abhängigkeit vom PREFERE-Studien Resultat (s. Flow Chart S. 6).

#### 7.3 Beschreibung des Studienablaufs

Nach der erfolgreichen Prüfung der Ein- und Ausschlusskriterien, dem erfolgten Patienten-Aufklärungsgespräch und der Unterschrift des Patienten auf der Einwilligungserklärung wird der Patient in einen der beiden Studienarme randomisiert.

#### 7.3.1 Randomisation

Die Randomisation wird vom ZKS Leipzig-KKS vorgenommen. Sie erfolgt nach dem Minimierungsalgorithmus nach Pocock (s. Kap. 9.1) im Verhältnis von R-LRPE zu LRPE von 3:1.

Die Randomisation der Patienten erfolgt bei der Baseline-Visite. Auf der Randomisationsanforderung an das ZKS-Leipzig-KKS bestätigt ein Prüfarzt, dass der Patient alle Einschlussund keine der Ausschlusskriterien für die Aufnahme in die Studie erfüllt.

Schrittfolge für den Randomsierungsvorgang

- 1. Fax des ausgefüllten Randomisationsformulars vom Prüfzentrum an das ZKS Leipzig-KKS (Mo-Fr. 8:00 h bis 17:00 h)
- 2. datenbankgestützte Randomisation im ZKS Leipzig-KKS
- 3. automatischer Faxversand des Randomisationsergebnisses an das Prüfzentrum

#### 7.3.2 Datenerhebung zur Baseline

- Zeitpunkt: stationäre Aufnahme zur radikalen Prostatektomie
- Prüfung der Ein- und Ausschlusskriterien
- Einwilligungserklärung nach erfolgter Aufklärung
- Ausführliche Anamnese
- Karnofsky-Performance-Status
- Randomisation
- Ausfüllen der Patientenfragebögen
  - ICIQ-SF
  - PAD-Verbrauch
  - IIEF-5
  - REF
  - EORTC QLQ-C30
  - EORTC QLQ-PR25
  - HADS
- Aktivitätslevel, Trinkmenge
- Begleitmedikation und Begleiterkrankungen (Quelldaten)
- PSA-Wert

#### 7.3.3 Chirurgischer Eingriff und perioperative Datenerhebung

Chirurgische Verfahren im Rahmen der Studie werden gemäß der Gebrauchsanweisung und/oder des Benutzerhandbuchs für das jeweilige Produkt durchgeführt.

Die zugewiesene Behandlungsmethode muss für die Entfernung der tumorbefallenen Prostata verwendet werden.

Dokumentation für den chirurgischen Eingriff und die peri- und frühe postoperative Phase (Quelldaten):

- Name des Chirurgen
- Eingriffsdauer
- Intraoperative Komplikationen
- Dauer der Katheterisierung
- Krankenhausliegedauer
- Klinische Daten (Tumorlokalisation, Tumorstadium, Gleason Score, Zugangsweg, Blutverlust, Transfusionen, Lymphadektomie, Prostatagewicht, Nerverhalt, Residualtumor)

Tabelle 3 Definition der Zeitmessung

| Messung | Zeitpunkt des Beginns | Zeitpunkt der Beendigung |
|---|---|---|
| Eingriffsdauer | Erster Schnitt für ersten Trokar | Nahtende |
| Dauer der Katheterisierung | Katheter wird eingeführt | Katheter wird entfernt <sup>1</sup> |
| Krankenhausliegedauer | Tag der stationären Aufnahme<br>(Tag vor OP) | Entlassungsdatum aus dem primären KH/von der primären Station |

<sup>&</sup>lt;sup>1</sup> In Ausnahmefällen ist eine erneute Katheterisierung notwendig, dann gilt als Endpunkt die Entfernung des letzten Katheters.

#### 7.3.4 Datenerhebung zu den Follow-up-Visiten

Tabelle 4 Zeitfenster für Nachbeobachtungstermine

| Nachbeobachtungstermin | Compliance-Fenster | Tage nach dem Eingriff |
|------------------------|-------------------------|------------------------|
| 1 Monat (30 Tage) | plus oder minus 10 Tage | 20-40 |
| 3 Monate (90 Tage) | plus oder minus 10 Tage | 80-100 |
| 6 Monate (180 Tage) | plus oder minus 20 Tage | 160-200 |
| 12 Monate (365 Tage) | plus oder minus 30 Tage | 335-395 |
| 24 Monate (730 Tage) | plus oder minus 60 Tage | 670-790 |
| 36 Monate (1095 Tage) | plus oder minus 60 Tage | 1035-1155 |

Zu den Follow-Up Visiten nach 1, 3, 6 und 12 Monaten werden Patientenfragebögen zusammen mit einem frankierten Rückumschlag versendet. Um die drop-out Rate gering zu halten, werden die Patienten vor jedem Follow-Up Zeitpunkt telefonisch kontaktiert. Bleiben Bögen aus, erfolgt in der Regel eine schriftliche oder telefonische Benachrichtigung des Patienten. Das Follow-Up Management (telefonische Kontaktierung, Versendung der Bögen, Dateneingabe) erfolgt durch die Studienzentrale in Leipzig.

#### Tag der Katheterentfernung bis 3 Monate postoperativ

Patienten-Tagebuch zu PAD-Verbrauch, Aktivitätslevel, Trinkmenge

#### 1 Monat postoperativ

- Patientenfragebögen:
  - ICIQ-SF
  - EORTC QLQ-C30
  - EORTC QLQ-PR25
  - HADS
  - Patientenzufriedenheit
- Begleitmedikation (Medikamente, die sich auf die Urogenitalfunktion auswirken)
- Erektionshilfen (potenzfördernde Medikamente, u. ä.)

#### 3 Monate postoperativ

- Patientenfragebögen
  - PAD-Verbrauch
  - ICIQ-SF
  - IIEF-5
  - REF
  - EORTC QLQ-C30
  - EORTC QLQ-PR25
  - HADS
  - Patientenzufriedenheit
- Aktivitätslevel, Trinkmenge

- Begleitmedikation (Medikamente, die sich auf die Urogenitalfunktion auswirken)
- Erektionshilfen (potenzfördernde Medikamente, u. ä.)
- PSA-Wert

#### 6 Monate postoperativ

- Patientenfragebögen
  - PAD-Verbrauch
  - ICIQ-SF
  - IIEF-5
  - REF
  - EORTC QLQ-C30
  - EORTC QLQ-PR25
  - HADS
  - Patientenzufriedenheit
- Aktivitätslevel, Trinkmenge
- Begleitmedikation (Medikamente, die sich auf die Urogenitalfunktion auswirken)
- Erektionshilfen (potenzfördernde Medikamente, u. ä.)
- PSA-Wert

#### 12 Monate postoperativ

- Patientenfragebögen
  - PAD-Verbrauch
  - ICIQ-SF
  - IIEF-5
  - REF
  - EORTC QLQ-C30
  - EORTC QLQ-PR25
  - HADS
  - Patientenzufriedenheit
- Aktivitätslevel, Trinkmenge
- Begleitmedikation (Medikamente, die sich auf die Urogenitalfunktion auswirken)
- Erektionshilfen (potenzfördernde Medikamente, u. ä.)
- PSA-Wert
- Abfrage adjuvanter Therapien, diagnostizierter Rezidive, Metastasen

#### 24 und 36 Monate postoperativ

- PSA-Wert
- Abfrage adjuvanter Therapien, diagnostizierter Rezidive, Metastasen

#### 7.3.5 Vorzeitiger Abbruch der Studientherapie oder der Nachbeobachtung

Patienten werden aus der Studie ausgeschlossen, wenn einer der folgenden Gründe eintritt:

- bei Protokollverletzungen, die eine weitere Studienteilnahme unmöglich machen
- durch ärztliche Entscheidung (Gefährdung Patientensicherheit)
- wegen Kontaktverlust
- bei Rückzug der Einwilligungserklärung.

Bei Abbruch müssen die Gründe/Umstände und der letzte Status dokumentiert werden. Selbst bei Ausschluss eines Patienten aus der Studie wird dieser nachbeobachtet und dokumentiert, sofern der Patient seine Einwilligung nicht zurückzieht.

#### 7.4 Datenerfassung

#### 7.4.1 Kontinenz: PAD-Verbrauch

Die Anzahl der verwendeten Vorlagen (PADs) pro Tag (24 Stunden) sowie das Aktivitätslevel des Patienten (UCLA, s.u.) und die tägliche Trinkmenge werden in den ersten drei postoperativen Monaten in Form eines Patiententagebuches erfasst. Dieses Vorgehen hat entscheidende Vorteile. Niemand kann den Erfolg und die Auswirkungen der Therapie auf die Kontinenz besser einschätzen als der Patient selbst. Aussagekräftig sind vor allem Angaben, die Rückschlüsse auf den kontinuierlichen Verlauf zulassen. Deshalb sind engmaschige Verlaufsdaten in Form von Eintragungen in das Tagebuch essentiell. Gesundheitliche Belange werden in der Regel weniger konkret wiedergegeben, wenn sich Patienten nur auf ihre Erinnerung verlassen oder punktuell zu nur einem Zeitpunkt ihren Zustand angeben sollen. Die regelmäßigen Eintragungen ins Patiententagebuch hingegen funktionieren wie ein Protokoll. Sie ermöglichen einen genauen Überblick über den Verlauf der Kontinenz des Patienten. Ein weiterer Vorteil ist der Tatbestand der Realisierbarkeit, eine tägliche Messung bei großen Patientenzahlen im Längsschnitt umsetzten und daher möglichst lückenlos abbilden zu können.

#### 7.4.2 Patienten-Fragebögen

Zusätzlich werden validierte, international bewährte Fragebögen eingesetzt, die entsprechend ihres Auswertungsmanuals gehandhabt werden. Alle Fragebögen sind selbstständig vom Patienten auszufüllen.

#### Kontinenz: ICIQ-SF

Der International Consultation on Incontinence Questionnaire - Short Form, ICIQ-SF (Range 0–21) dient der Erfassung der Kontinenz. Ein entscheidendes Auswahlkriterium für seine Nutzung ist u.a., dass es ein national und international häufig eingesetztes Instrumentarium zur Messung von Kontinenz ist, welches am PAD-Test validiert ist (Twiss et al. 2007). Es findet zudem bei der Evaluation im Rahmen von Prostatakarzinomzentren (DKG) breite Anwendung.

#### **Erektile Funktion: IIEF-5**

Zur Erfassung der erektilen Dysfunktion wird der International Index of Erectile Function (IIEF-5) genutzt, der auch unter dem Namen Sexual Health Inventory for Men (SHIM) bekannt ist. SHIM enthält die 5 IIEF Fragen der Langversion (IIEF-15) mit dem höchsten diagnostischen Vorhersagewert für erektile Dysfunktion (Rosen et al. 1999). Eine Validierungsstudie der deutschsprachigen IIEF-Version wurde 2003 von Wiltink et al. vorgelegt. Die fünf Items des SHIM trennen gut zwischen Männern mit und ohne erektile Dysfunktion (ED) und reflektieren den Schweregrad der ED (Kategorisierung der ED: keine ED (≥ 22), mild (16-21), moderate (11-15) und schwer (<11).

#### Aktivitätslevel: UCLA

Die Erfassung des individuellen Aktivitätsniveaus erfolgt in Anlehnung an das 10-Punkte Activity-Level Rating der University of California Los Angeles (Zahiri et al. 1998). Die Einteilung richtet sich danach, welche Anstrengung im Alltag bzw. welche sportlichen Aktivitäten der Patient leistet. Der Score weist zehn verschiedene Aktivitätsstufen auf. Der Patient ordnet sich selbst entsprechend der Skala einem Level zu. Die Abstufung reicht dabei von absolut inaktiv (Level 1) über moderate Aktivitäten wie regelmäßige Teilnahme an Arbeiten im Haus/Garten und gelegentlichem Freizeitsport (Level 5 - 6), bis hin zu regelmäßiger sportlich anspruchsvoller Aktivität (Level 10). Je niedriger das Level, umso geringer sind jeweils die

Aktivitäten, die vom Patienten durchgeführt werden. Gerade für das hier zu untersuchende ältere Patientenkollektiv ist eine Einteilung nach dem UCLA-Rating sehr gut geeignet.

#### Gesundheitsbezogene Lebensqualität: EORTC QLQ-C30

Die Lebensqualitätsdaten werden mit den validierten und international anerkannten Lebensqualitätsfragebögen der EORTC (European Organization for Research and Treatment of Cancer) erfasst. Der EORTC QLQ-C30 (Quality of Life Questionnaire - Core 30) wurde speziell zur Messung der gesundheitsbezogenen Lebensqualität von Krebspatienten entwickelt (Aaronson et al., 1993). Die 30 Items des Instruments umfassen fünf Funktionsskalen (körperliche, Rollen-, emotionale, kognitive und soziale Funktion), drei Symptomskalen (Fatigue, Schmerz, Übelkeit), sechs Einzelitem-Skalen (Schlafstörungen, Kurzatmigkeit, Durchfall, Appetitlosigkeit, Verstopfung, finanzielle Schwierigkeiten) sowie eine globale Gesundheits-/Lebensqualitätsskala. Ein weiterer Vorteil der EORTC Bögen besteht im Vorliegen repräsentativer Referenzdaten, die von der Allgemeinbevölkerung und verschiedenen Indikationen vorliegen. Der QLQ-C30-Basisbogen kann ergänzt werden durch die krankheitsspezifischen EORTC-Module (u.a. EORTC QLQ-PR25).

#### Prostataspezifische Lebensqualität: EORTC QLQ-PR25

Der EORTC QLQ-PR25 evaluiert spezifische Belastungen und Probleme von Prostatakarzinompatienten (van Andel et al. 2008). Er umfasst zwei Funktionsskalen (sexuelle Aktivität und sexuelle Funktion), drei Symptomskalen (Blasen-, Darm- und behandlungsbezogene Symptome) und eine Single-Item-Skala zur Messung der Belastung durch Inkontinenzhilfen. Die der Psychoonkologie entstammenden EORTC-Bögen erweitern die oben genannten Fragebögen zur Kontinenz und erektilen Funktion (IIEF und ICIQ) um eine stärker psychosoziale Komponente und stellen das Gesamtbefinden und die subjektive Wahrnehmung des Patienten in den Mittelpunkt.

Die EORTC-Fragebögen werden entsprechend des EORTC Auswertungsmanuals verwendet (Fayers et al. 1995). Alle Skalenwerte werden linear transformiert auf einer 0-100 Punkteskale. Höhere Werte auf einer Funktionsskala repräsentieren eine bessere Funktion/Lebensqualität. Dagegen zeigen höhere Werte auf einer Symptomskala eine stärkere Symptomlast an. Basierend auf bisherigen Forschungsergebnissen wird eine Differenz von 10 und mehr Punkten zwischen zwei Zeitpunkten oder zwischen zwei Gruppen als klinisch relevant betrachtet (King 1995; Osoba et al. 1998; Pietrow et al. 2001; Rodrigues et al. 2004).

#### **Psychisches Befinden: HADS**

Zur Erfassung von Ängstlichkeit und Depressivität wird die deutsche Version der Hospital Anxiety and Depression Scale (HADS) verwendet (Hermann et al. 1995). Sie besteht aus einer Angst- und einer Depressivitätsskala und wurde für Patienten mit primär körperlichen Erkrankungen konzipiert. Anhand von Cut-off Werten ist eine Fallidentifikation möglich.

#### Residuale Erektile Funktion: REF

Die Beurteilung der "Residual Erectile Function" basiert auf dem validierten, Single-Item "Erection Hardness Score (EHS)", wie von Mulhall et al. 2007 beschrieben. Sie wird auf der Grundlage der individuellen Angabe des Patienten vorgenommen.

Der Score ist ein gut geeigneter Parameter für den Erfolg einer Therapie. Anhand des EHS, der von dem US-Urologen Erwin Goldstein nach klinischen Erfahrungen und dem subjektiven Empfinden der Patienten entwickelt worden ist, werden verschiedene Härtegrade von Erektionen unterschieden. Hierbei soll der Patient den Härtegrad seiner Erektion auf einer 5-Punkteskala von 0 (Penis hat sich nicht vergrößert) bis 4 (Penis ist komplett hart und völlig steif) angeben.

#### Patientenzufriedenheit mit der chirurgischen Behandlung

Probanden werden zu hinsichtlich ihrer Zufriedenheit mit der chirurgischen Behandlung befragt, um ihre Wahrnehmung des Verfahrens und der postoperativen Erholung zu beurteilen (z. B. Annehmlichkeit des Verfahrens, Wirksamkeit, Tolerierbarkeit der Nebenwirkungen und Erholungsdauer, Rückkehr ins Arbeitsleben).

#### 7.4.3 Klinische Daten

Klinische Daten werden der klinikinternen Dokumentation (Quelldaten) entnommen. Die Erfassung der Komplikationen erfolgt einheitlich gemäß der Clavien Klassifikation, einem standardisierten Verfahren zur Erfassung negativer chirurgischer Ergebnisse (Clavien et al. 2009, Dindo et al. 2004, Stolzenburg et al. 2006). Unterschieden werden hierbei OP-Komplikationen, Früh- (<1 Monat p.o.) und Spätkomplikationen (> 1 Monat p.o.).

Quelldaten sind Originalinformationen zum Patienten und befinden sich in Quelldokumenten. Beispiele für Originaldokumente und -datensätze dieser Art sind: Krankenhausunterlagen (papierbasiert oder elektronisch), Klinik- und Praxisdiagramme, Laborergebnisse, Memoranden, Patientenfragebögen, Patiententagebücher oder Bewertungschecklisten, Rezepturunterlagen von Apotheken, Datenaufzeichnungen automatisierter Instrumente, nach Verifikation als richtig und vollständig beglaubigte Kopien oder Transkriptionen, Röntgenaufnahmen, Patientenakten sowie Aufzeichnungen in Labors und medizintechnischen Abteilungen, die an der klinischen Studie beteiligt sind. Für jeden Patienten müssen sämtliche die Studie betreffenden Quelldaten zwingend vorliegen. Im Rahmen der Datenschutzerklärung muss sichergestellt werden, dass klinische Monitore, Auditoren und Inspektoren Einsicht in die Quelldaten nehmen dürfen.

#### 7.4.4 Onkologische Daten

Die Erfassung des PSA-Wertes sowie einer ggf. adjuvanten Therapie und diagnostizierter Rezidive und Metastasen erfolgt in einer längsschnittlichen Perspektive bis 3 Jahre postoperativ. Der PSA-Wert wird im Rahmen der Prostatektomie-Nachsorge regelmäßig durch den niedergelassenen Urologen erhoben (im ersten postoperativen Jahr aller drei Monate; im zweiten und dritten postoperativen Jahr halbjährig). Nach radikaler Prostatektomie kennzeichnet ein in mindestens zwei Messungen bestätigter PSA-Wert >0,2 ng/ml ein biochemisches Rezidiv (siehe S3-Leitlinie der DGU 2011). Die PSA-Wert Bestimmung erfolgt im Rahmen der Prostatektomie-Nachsorge, PSA-Laborbefunde werden mit Angabe des Herstellers und der Methode (Testkit) auf Grundlage der Referenzwerte dokumentiert.

#### 7.4.5 Medikamente

Informationen über Medikamente, die der Patient zum Zeitpunkt des Visitentermins einnimmt und die sich auf Urogenitalfunktion auswirken oder auf die Erektionsfähigkeit (sog. erektionsfördernde Hilfsmittel, z.B. Viagra) werden vom Baseline-Termin bis zum 12 Monats-Follow-Up erfasst.

#### 7.5 Vorzeitiger Abbruch für Studienpatienten

Einer oder mehrere der folgenden Umstände können zu einem Abbruch der Studie bei einem einzelnen Patienten führen:

- Rücknahme der Einwilligung des Patienten
- Verletzung des Studienprotokolls, sofern diese eine Weiterbehandlung unmöglich macht
- Nachträgliches Bekanntwerden/ Auftreten eines Ausschlusskriteriums, sofern es eine Weiterbehandlung unmöglich macht

## 8 Unerwünschte Ereignisse (AE/SAE/Vorkommnis)

#### 8.1 Unerwünschtes Ereignis - AE

#### 8.1.1 Definition

Unerwünschte Ereignisse sind alle bei Versuchspersonen, dem Anwender oder bei anderen Personen auftretenden unerwünschten medizinischen Ereignisse, unbeabsichtigte Erkrankungen oder Verletzungen oder unerwünschte klinische Diagnosen (inkl. abnormer Laborergebnisse) egal, ob diese in kausaler Beziehung zu dem Medizinprodukt stehen oder nicht.

Diese Definition schließt Ereignisse im Zusammenhang mit dem Medizinprodukt oder dem Vergleichsprodukt und den beteiligten Verfahren ein.

Für Anwender oder andere Personen ist diese Definition auf Ereignisse im Zusammenhang mit dem Medizinprodukt beschränkt.

Definition ISO 14155: 2012-01.

#### 8.1.2 Dokumentation und Meldung

Alle AEs werden auf dem AE-Bogen des CRFs und in der Patientenakte zusammen mit der eventuell angewendeten Begleitmedikation dokumentiert. Hierbei werden die Diagnose, Beginn und Ende, Schweregrad, möglicher kausaler Zusammenhang mit der Prüftherapie und Ausgang des Ereignisses dokumentiert. Der Prüfarzt verfolgt den Verlauf des Ereignisses, bis das AE beendet ist oder der Patient stabilisiert ist.

AEs werden für die Zeit der Krankenhausbehandlung erfasst sowie im Rahmen der regelmäßigen Nachsorge der Patienten (Krebsscreening nach der Operation) für eine maximale Dauer von 36 Monaten (Ende der Nachbeobachtung) nach der Intervention abgefragt.

Bei einem AE, das nicht durch die unter 8.2.1 beschriebenen Kriterien zu einem SAE wird, bestehen keine besonderen Meldepflichten.

#### 8.2 Schwerwiegendes unerwünschtes Ereignis (SAE)

#### 8.2.1 Definition

Ein unerwünschtes Ereigniss wird laut Medizinproduktesicherheitsplanverordnung (MPSV §2 und ISO 14155: 2012-01) als schwerwiegend definiert, wenn es:

- a) zum Tod führte,
- b) zu einer schweren Gesundheitsbeeinträchtigung der Versuchsperson führte, die entweder
  - 1) eine lebensbedrohende Erkrankung oder Schädigung zur Folge hat, oder
  - 2) eine dauernde Beeinträchtigung einer Körperstruktur oder -funktion zur Folge hat, oder

- 3) die Krankenhausaufnahme oder die Verlängerung eines bestehenden Krankenhausaufenthaltes zur Folge hat, oder
- 4) einen medizinischen oder chirurgischen Eingriff zur Folge hat, um eine lebensbedrohende Krankheit oder Verletzung oder eine dauernde Beeinträchtigung einer Körperstruktur oder -funktion zu verhindern,
- c) zur Schädigung eines Fetus, zum Fetaltod, einer kongenitalen Fehlbildung oder einem Geburtsschaden führte.

ohne zu berücksichtigen, ob das Ereignis vom Medizinprodukt verursacht wurde.

Anmerkung: Ein geplanter Krankenhausaufenthalt auf Grund vorher vorhandener Gegebenheiten oder ein vom CIP gefordertes Verfahren, ohne eine beträchtliche Verschlechterung des Gesundheitszustandes wird nicht als schwerwiegendes unerwünschtes Ereignis betrachtet.

#### 8.2.2 Dokumentations- und Meldeverpflichtungen für den Prüfer

Eine Meldung von SAEs an die Bundesoberbehörde ist nicht erforderlich, da diese Studie nach §23b MPG durchgeführt wird. Sollten seitens einer nach Berufsrecht zuständigen Ethikkommission SAE- und/oder Vorkommnismeldungen bestehen, so wird diesen nachgekommen.

Aufgetretene SAEs werden durch den Prüfer auf den SAE-Bögen dokumentiert und im Rahmen der Endauswertung analysiert.

Hinweise zum Ausfüllen des Formblattes finden sich in einer entsprechenden Working Instruction für den Prüfer, welche im Investigator Site File vorliegt.

#### 8.3 Vorkommnis

#### 8.3.1 Definition

Gemäß §29 (1) MPG ist ein Vorkommnis:

- jede Funktionsstörung, jeder Ausfall oder jede Änderung der Merkmale oder der Leistung eines Medizinproduktes sowie jede Unsachgemäßheit der Kennzeichnung oder Gebrauchsanweisung, die direkt oder indirekt zum Tod oder zu einer schwerwiegenden Verschlechterung des Gesundheitszustandes eines Patienten oder eines Anwenders oder einer anderen Person geführt haben oder hätten führen können,
- jeden Grund technischer oder medizinischer Art, der auf Grund der in Nummer 1 genannten Ursachen durch die Merkmale und die Leistungen eines Medizinproduktes bedingt ist und zum systematischen Rückruf von Medizinprodukten desselben Typs durch den Hersteller geführt hat.

Eine schwerwiegende Verschlechterung des Gesundheitszustands kann folgendes umfassen:

- a) Lebensbedrohende Krankheit (oder Verletzung);
- b) dauerhafte Beeinträchtigung einer Körperfunktion oder dauerhafter Körperschaden
- c) ein Zustand, der eine medizinische oder chirurgische Intervention erfordert, um a) oder b) zu vermeiden (z.B. klinische relevante Verlängerung der Dauer einer Operation; Erfordernis einer Krankenhausbehandlung oder wesentliche Verlängerung eines Krankenhausaufenthalts);

d) Eine indirekte Schädigung [...] als Folge eines fehlerhaften Ergebnisses einer diagnostischen oder labordiagnostischen Untersuchung, wenn die Produkte gemäß der Gebrauchsanweisung des Herstellers angewendet wurden; Gefährdung oder Tod eines ungeborenen Kindes, jegliche angeborene Anomalie oder Geburtsschäden.

#### 8.3.2 Meldeverpflichtungen für den Prüfer

Vorkommnisse werden

- auf dem dafür vorgesehenen Vorkommnis-Formblatt dokumentiert und
  - müssen unverzüglich an die Bundesoberbehörde (BfArM) gemeldet werden. Zur Meldung an das BfArM steht auf der Webseite des BfArM ein "Formblatt für die Meldung von Vorkommnissen durch sonstige Inverkehrbringer sowie Betreiber und Anwender nach §3 Abs. 2 bis 4 der Medizinprodukte-Sicherheitsplanverordnung" zur Verfügung.

#### 8.4 Sicherheitsanalysen

Im Rahmen der Studie sind keine gesonderten Sicherheitsanalysen notwendig, da das Sicherheitsprofil der verwendeten Techniken etabliert ist und die Patienten eine Regelbehandlung erfahren.

Jeder Patient wird hinsichtlich der Sicherheit im Studienverlauf engmaschig überwacht. Dies beinhaltet die Erfassung von unerwünschten Ereignissen für die Zeit des primären Krankenhausaufenthaltes sowie die regelmäßige Nachuntersuchung mit onkologischer Verlaufskontrolle (PSA-Wert).

#### 8.5 Begleiterkrankungen

Begleiterkrankungen, die kein Ausschlusskriterium darstellen, werden zu Beginn der Studie dokumentiert und im Rahmen der Studienuntersuchungen evaluiert. Es wird keine Verschlechterung von Begleiterkrankungen durch die Studientherapie erwartet. Sollte dies dennoch auftreten, oder eine neue Begleiterkrankung während der Studienteilnahme diagnostiziert werden, muss der behandelnde Prüfarzt dies auf dem CRF dokumentieren sowie beurteilen, ob dies ein Grund für einen Studienabbruch sein könnte.

#### 8.6 Therapeutische Maßnahmen

Bedarf der Patient aufgrund des unerwünschten Ereignisses einer Behandlung, so muss diese nach dem derzeitigen Stand der medizinischen Forschung durchgeführt werden, um die Gesundheit des Patienten wieder herzustellen. Geeignete Geräte und Präparate zur Wiederbelebung müssen verfügbar sein, um den Patienten im Notfall schnellstmöglich behandeln zu können.

Die Behandlung des AE bzw. SAE muss dokumentiert werden.

Die ergriffenen Maßnahmen müssen vom Prüfarzt entweder an der entsprechende Stelle im CRF und/oder durch zusätzliche Unterlagen dokumentiert werden

- Behandlung unterbrochen
- Behandlung nicht unterbrochen
- unbekannt
- nicht zutreffend

#### 8.7 Korrektive Maßnahmen

Korrektive Maßnahmen sind Maßnahmen zur Beseitigung, Verringerung oder Verhinderung des erneuten Auftretens eines von einem Medizinprodukt ausgehenden Risikos (§2, Abs. 2 MPSV).

Treten während der klinischen Prüfung Umstände auf, die die Sicherheit der Patienten, Anwender oder Dritter beeinträchtigen können, so ergreifen die Studienleitung sowie die die klinische Prüfung durchführenden Personen unverzüglich alle erforderlichen Sicherheitsmaßnahmen, um die Patienten, Anwender oder Dritte vor unmittelbarer oder mittelbarer Gefahr zu schützen. Die ergriffenen Maßnahmen müssen vom Prüfarzt entweder an der entsprechenden Stelle im CRF und/oder durch zusätzliche Unterlagen dokumentiert werden.

#### 8.8 Klassifikation unerwünschter Ereignisse

#### 8.8.1 Schweregrad

Der Schweregrad eines unerwünschten Ereignisses wird entsprechend der Definitionen im Kapitel 8.1 und 8.2 beurteilt.

#### 8.8.2 Beurteilung der Intensität

Die Beurteilung der Intensität erfolgt entsprechend der CTCAE V3.0.

| | Leichtes Ereignis keine spezielle medizinische Intervention notwendig, |
|---|---|
| Mild Adverse<br>Event | <ul> <li>ausschließlich asymptomatische Laborergebnisse oder Röntgen-<br/>befunde,</li> </ul> |
| | <ul> <li>geringe medizinische Relevanz</li> </ul> |
| Moderate Ad-<br>verse Event | <ul> <li>Moderates/mittelschweres Ereignis</li> <li>minimale medizinische Intervention erforderlich bzw. Intervention lokal begrenzt,</li> </ul> |
| | <ul> <li>ausschließlich nichtinvasive Maßnahmen (z.B. Wickel) notwendig</li> </ul> |
| Severe and un-<br>desirable Ad-<br>verse Event | Schweres und nicht erwünschtes Ereignis <ul> <li>signifikante Symptome, die einen Krankenhausaufenthalt oder invasive Interventionen erfordern,</li> </ul> |
| | <ul> <li>z.B. Transfusionen, elektive interventionelle radiologische Maß-<br/>nahmen, therapeutische Endoskopie oder Operation</li> </ul> |
| Life-threatening<br>or disabling<br>Adverse Event | Lebensbedrohliches oder zur Behinderung führendes Ereignis verschärft durch akute, lebensbedrohliche Komplikationen des Stoffwechsels oder des Kreislaufsystems, z.B. Kreislaufkollaps, Hämorrhagie, Sepsis |
| | <ul> <li>lebensbedrohliche physiologische Konsequenzen,</li> </ul> |
| | <ul> <li>Notwendigkeit intensiver Betreuung, umgehender invasiver, interventioneller oder radiologischer Maßnahmen, therapeutische Endoskopie oder Operation</li> </ul> |
| Death related to<br>Adverse Event | Tod als Folge des AE |

#### 8.8.3 Beurteilung des Kausalzusammenhanges

Der Prüfer muss beurteilen, ob seiner Meinung nach das Auftreten des unerwünschten Ereignisses in einem kausalen Zusammenhang mit der Anwendung des Prüfprodukts steht. Dabei ist die unten genannte Klassifikation anzuwenden. Jedes unerwünschte Ereignis muss dokumentiert werden, auch wenn kein Zusammenhang mit der Anwendung des Prüfprodukts zu erkennen ist.

- Möglich
- Nicht Möglich

Als **Möglich** wird der Zusammenhang bewertet, wenn eines der folgenden Kriterien nach WHO-UMC erfüllt ist:

- plausibler zeitlicher Zusammenhang, und kann nicht durch Begleiterkrankung oder andere Produkte erklärt werden, und positive Reaktion auf Absetzen, und bekannte pharmakologische oder phänomenologische Reaktion und positive Wiedergabe des Produktes, wenn notwendig
- Begründeter zeitlicher Zusammenhang, und Erklärung durch Begleiterkrankung oder andere Produkte unwahrscheinlich, und Positive Reaktion auf Absetzen
- Begründeter zeitlicher Zusammenhang, aber Erklärung durch andere Produkte oder Begleiterkrankung möglich, Informationen über Absetzen sind unvollständig oder unklar
- Weitere Informationen notwendig, um Beurteilung exakt vorzunehmen
- Beurteilung nicht möglich, da die Informationen unzureichend oder widersprüchlich sind

Als **Nicht Möglich** wird der Zusammenhang bewertet, wenn das folgende Kriterium nach WHO-UMC erfüllt ist:

Zeitlicher Zusammenhang macht den kausalen Zusammenhang unwahrscheinlich, **und** andere Produkte oder zugrunde liegende Erkrankungen liefern plausible Erklärung

Eine unerwünschte Wirkung (Adverse Device Effect, ADE) des Medizinproduktes (ISO 14155-1:2003, Punkt 3.1) ist ein dem Medizinprodukt zuzuschreibendes, unerwünschtes Ereignis. Eine unerwünschte Wirkung des Produktes, die zu einer der Folgen führte, die für ein schweres unerwünschtes Ereignis kennzeichnend sind oder die zu einer dieser Folgen geführt hätten, wenn keine geeigneten Maßnahmen ergriffen worden wären, nicht dagegen eingeschritten worden wäre oder wenn die Umstände weniger günstig gewesen wären entspricht einem Serious Adverse Device Effect (SADE) (EN ISO 144155-1:2012-01).

Anmerkung 1: Diese bezieht unerwünschten Ereignisse ein. die sich aus nicht ausreichenden oder ungenauen Anleitungen für den Gebrauch, die Aufstellung, die Implantation, die Installation. oder das Funktionieren oder etwaige Fehlfunktionen des Prüfproduktes ergeben.

Anmerkung 2: Dies bezieht alle Ereignisse ein, die auf einen Benutzungsfehler oder auf einen bewussten Fehlgebrauch des Prüfprodukts zurückzuführen sind.

#### 8.8.4 Erwartet / Unerwartet

Unerwartet sind unerwünschte Ereignisse dann, wenn sie nicht in der aufgetretenen Art oder in der aufgetretenen Intensität im Handbuch des Prüfers oder im Prüfplan beschrieben sind.

Eine unvorhersehbare schwerwiegende unerwünschte Wirkung des Produkts (unanticipated serious adverse device effect/USADE) entspricht einer schwerwiegenden unerwünschten Wirkung des Produkts. die wegen ihrer Art, ihres Auftretens, der Schwere oder der Folgen in der aktuellen Version im Handbuch des Prüfers oder im Prüfplan nicht beschrieben ist.

#### 8.8.5 Ausgang des unerwünschten Ereignisses

Der Ausgang eines unerwünschten Ereignisses wird wie folgt klassifiziert:

- wiederhergestellt
- wiederhergestellt mit Folgeschäden
- fortbestehend
- tödlich \*
- unbekannt

\*Achtung: Der Tod eines Patienten ist an sich kein Ereignis, sondern dessen Ergebnis. Das Ereignis, welches zum Tod des Patienten geführt hat, muss vollständig dokumentiert und gemeldet werden, auch wenn der Tod erst vier Wochen nach Ende der Studienbehandlung / Anwendung des Medizinproduktes aufgetreten ist und unabhängig davon, ob es einen Zusammenhang mit der Therapie gibt oder nicht.

#### 9 Biometrie

#### 9.1 Randomisationsalgorithmus

Patienten werden mit Hilfe des Pocock-Optimierungsverfahrens (Pocock and Simon 1975) im Verhältnis 3 : 1 (R-LRPE vs. LRPE) randomisiert. Das Rando-Verhältnis R = 3 (und damit eine 3/4-Chance, durch das neue, innovativere Verfahren behandelt zu werden) soll Patienten zur Studienteilnahme motivieren.

Bei der datenbankgestützten Randomisierung werden folgende Strata berücksichtigt:

- A1: nicht nerverhaltend, A2: einseitig nerverhaltend, A3: zweiseitig nerverhaltend,
- B1: Alter ≤ 65, B2: Alter > 65
- C: Studienzentrum (C1 ... C4)

#### 9.2 Endpunkte der Studie

#### 9.2.1 Primärer Endpunkt

Primärer Endpunkt ist die Zeit bis zum Erreichen der Kontinenz (bis 3 Monate postoperativ). Dazu wird der tägliche Bedarf an PADs erfasst. Ein Patient gilt dann als kontinent, wenn er an drei aufeinanderfolgenden Zeitpunkten keine PADs mehr benötigt hat. Diese Definition von Kontinenz als binäres Merkmal ist vergleichbar mit dem Kriterium ICIQ=0, welches die DKG im Rahmen der Evaluation von Prostatakarzinomzentren empfiehlt. So ermöglicht dieser relativ "harte" Endpunkt den Vergleich mit anderen Methoden in der Literatur.

Die Analyse der "Zeit-bis-Ereignis-Daten" hat den weiteren Vorteil, dass Patienten, welche vorfristig die Studie verlassen, nicht aus der Analyse heraus fallen, sondern die Zeiten bis zum Studienende gelten im Sinne der Überlebenszeitanalyse als "zensiert".

#### 9.2.2 Sekundäre Endpunkte

Folgende Parameter werden, wenn nicht anders angegeben, jeweils nach 1, 3, 6 und 12 Monaten ausgewertet:

 Kontinenz (ICIQ-SF-Score, Anzahl verbrauchter PADs, Urinary Symptom Scale des EORTC QLQ-PR25) <u>Hinweis</u>: In der Literatur sind die Korrelationen zwischen den verschiedenen Kontinenzmaßen wenig untersucht bzw. dokumentiert. Die Erfassung und Auswertung von PAD-Verbrauch und ICIQ-Score kann helfen, diese Lücke zu verkleinern.

- Erektile Funktion (IIEF-5) nach 3, 6, 12 Monaten p.o.
- Residuale Erektile Funktion (REF) nach 3, 6, 12 Monaten p.o.
- Gesundheitsbezogene Lebensqualität (EORTC QLQ-C30)
- Prostataspezifische Lebensqualität (EORTC QLQ-PR25)
- Angst und Depressivität (HADS)
- Patientenzufriedenheit
- PSA-Wert nach 3, 6, 12, 24, 36 Monaten
- perioperative Parameter (Blutverlust, Transfusionsrate, OP-Zeit, Komplikationen)
- Veränderung von ICIQ, IIEF, HADS und Lebensqualität im zeitlichen Verlauf
- Einflussfaktoren der Kontinenz

#### 9.3 Statistische Formulierung der Studienfrage

#### 9.3.1 Statistische Hypothese der primären Fragestellung

- $H_0$ : Die Zeit bis zum Erreichen der Kontinenz unterscheidet sich nicht zwischen LRPE- und R-LRPE-Patienten:  $t_{R-l,RPE} = t_{l,RPE}$
- $H_A$ : R-LRPE-Patienten werden schneller / langsamer kontinent als LRPE-Patienten.  $t_{R-LRPE} \neq t_{LRPE}$  (zweiseitige Fragestellung)

#### 9.4 Fallzahldiskussion

#### 9.4.1 Abschätzung der Effektgrößen

Der Behandlungseffekt wird daran gemessen, wie viele Patienten der R-LRPE-Gruppe eher kontinent werden als jene nach LRPE. Betrachtet man einen konkreten Zeitpunkt (3 Monate), so spiegelt sich dieser Unterschied als Differenz in Ereignisraten wider. Bisherige Studien zur Inkontinenz nach radikaler Prostatektomie kommen zu sehr unterschiedlichen Ergebnissen. Dokumentierte Kontinenzraten drei Monate postoperativ reichen von 17% bis 94% (Link et al. 2005; Berryhill et al. 2008; Ficarra et al. 2009; Kang et al. 2010). Diese Unterschiede dürften zum einen in unterschiedlichen soziodemographischen und medizinischen Merkmalen der Studienteilnehmer sowie unterschiedlichen Kriterien der Kliniken und Operateure begründet sein. Zum anderen spielen differente Methoden bei der Messung von Inkontinenz eine bedeutende Rolle (Boergermann et al. 2010). So weisen Studien, die Inkontinenz mit standardisierten Fragebögen messen, durchschnittlich niedrigere postoperative Kontinenzraten auf als Studien, bei denen der Kontinenzstatus des Patienten vom Arzt eingeschätzt wird (Herrman et al. 2007). Darüber hinaus gelten in verschiedenen Studien Patienten als komplett kontinent, die innerhalb von 24 Stunden bis zu eine Vorlage benötigen (auch bezeichnet als "sozial kontinent") (Boergermann et al. 2010). Nach Murphy (2010) verschleiern Begriffe wie "socially dry" und "security liner" den Sachverhalt und machen Vergleiche fast unmöglich.

Hinzu kommt, dass die Erfolgsaussichten nach nerverhaltender Operation deutlich besser sind als nach nicht-nerverhaltender Prostatektomie. Das verringert den zu erwartenden Behandlungseffekt für diese Untergruppe (mehr als 50% aller Patienten).

Für das Universitätsklinikum Leipzig liegen (noch unveröffentlichte) Pilotdaten zu den ersten 100 R-LRPE-Patienten vor. Dazu wurden aus 208 im gleichen Zeitraum herkömmlich laparoskopisch Operierten (LRPE) 100 Patienten nach Alter und nerverhaltender OP (s. 9.1) im
Verhältnis 1:1 gematcht. Demselben Ansatz folgten Hakimi et al. (2009), wo Paare von 75 R-LRPE-Patienten mit passenden herkömmlich laparoskopisch Operierten gebildet wurden. Beide Studien haben außerdem gemeinsam, dass in ihnen das strenge Kriterium für Kontinenz "no leakage, no pad" angewandt wurde.

In der Studie von Hakimi et al. wurden 3-Monats-Kontinenzraten von 54.6% (LRPE) bzw. 65.3% (R-LRPE) erzielt. Die Anteile jener Leipziger Patienten, von denen bereits das 3-Monats-Follow-up vorlag, liegen deutlich niedriger: LRPE 16/41 = 28%, R-LRPE: 15/34 = 44%. Das ist auch darauf zurückzuführen, dass hier fast 40% nicht nervschonend operiert werden mussten. Anhand dieser Daten liegt der Behandlungseffekt zwischen ~10 und 16%.

#### 9.4.2 Statistische Fehlergrößen

Die Irrtumswahrscheinlichkeit wird auf  $\alpha$  = 5% festgelegt. Für den Test des primären Endpunkts wird eine Power 1- $\beta$  = 80% angestrebt.

#### 9.4.3 Drop-outs

Patienten, bei denen sich nachträglich herausstellt, dass eine LRPE / R-LRPE nicht durchgeführt werden kann sowie Patienten, bei welchen nach der Randomisierung ein Tumorstadium 4 festgestellt wird, werden durch andere Patienten ersetzt. Sonst sind keine Ersetzungen vorgesehen.

Aufgrund des zweistufigen Rekrutierungsmodells (1. PREFERE, 2. LAP-01) wird geschätzt, dass etwa 40% der Patienten an der Studie teilnehmen.

Sowohl innerhalb der ersten drei Monate als auch zwischen 3. und 12. Monat werden je 10% Drop-outs erwartet (s. 4.3).

#### 9.4.4 Fallzahl- und Powerkalkulation

Der primäre Endpunkt soll mit dem Logrank-Test ausgewertet werden. Für Patienten, die aus der Studie ausscheiden, geht für die Analyse des primären Endpunkts die Zeit bis zu ihrem Studienende als zensierte Zeit in die Analyse ein. Die Studie wird anhand der Anteile ("proportions") von Patienten geplant, welche 3 Monate nach OP Kontinenz erreichen. Ausgangsbasis ist dabei eine Differenz der Kontinenzraten von 10% bei einem Anteil von 44% in der R-LRPE-Gruppe.

Da eine Zwischenauswertung vorgesehen ist, muss die Fallzahl für ein Gruppensequentielles Design berechnet werden. Die Statistiksoftware PASS (Hintze 2008) PASS 2008. NCSS, LLC. Kaysville, Utah) kalkuliert die Abbruchgrenzen anhand der von Jenisson & Turnbull (2000) empfohlenen Alpha-sparenden Methode nach Kim & deMets (vgl. auch 9.6). Bei 10% Drop-outs bis 3 Monate ergibt sich folgende Fallzahl:

Tabelle 5 Fallzahl

| N | LRPE | R-LRPE | P1 | P2 | HR | Diff | Power |
|-----|------|--------|-----|-----|-------|------|-------|
| 782 | 196 | 586 | 34% | 44% | 0.717 | 0.10 | 0.80 |

P1, P2: Anteile nach 3 Monaten kontinenter Patienten, HR: Hazard Ratio, Diff: Differenz der Anteile (= Behandlungseffekt)

Die Software PASS berechnet für den Fall balancierter Arme 292 notwendige Events. Durch das Umrechnen auf das Armverhältnis 3:1 ergeben sich die obigen Fallzahlen (Tab. 5). Dabei sind 10% Drop-outs bis 3 Monate bereits mit einkalkuliert. Es ist wahrscheinlich, dass ein Teil der Patienten, welche bis 3 Monate die Studie verlassen, informativ für die Analyse sind.

Das jährliche Aufkommen von Studienpatienten in den vier Zentren wird auf ca. 300 Patienten geschätzt (vgl. 4.3). Um die Fallzahl N = 782 Patienten zu erreichen, sollte 3 Jahre rekrutiert werden. Dadurch bleibt noch ein Prozentsatz für den Ersatz von Patienten (s. 9.4.3).

Das konservative Herangehen bei der Fallzahlschätzung dürfte dazu führen, dass die Studie für die Untersuchung vieler sekundärer Endpunkte (z. B. der ICIQ-Score als metrische Größe) sehr gut gepowert ist. Außerdem erlaubt die relativ hohe Fallzahl die Analysen von Subgruppen wie z. B. nerverhaltende vs. nicht-nerverhaltende OP.

# 9.5 Verfahren zur Datenanalyse

#### 9.5.1 Geplante Analysemethoden

Die Analyse erfolgt auf Intention-to-Treat- (ITT-)Basis, d. h. alle randomisierten Patienten, welche mit LRPE bzw. R-LRPE operiert wurden, gehören zur Auswertungspopulation.

Die Studienkohorte wird durch Mittelwert und Standardabweichung für kontinuierliche Größen, Anzahl und Prozent für qualitative Größen beschrieben. Extreme Abweichungen von der Normalverteilung werden anhand von Histogrammen erkannt. Für diese Größen ist die Beschreibung durch Median [Interquartile Range] geeignet.

Die Zeit bis zum Erreichen von Kontinenz bis 3 Monate nach Operation wird durch (inverse) Kaplan-Meier-Kurven dargestellt und mit dem Logrank-Test verglichen. Mittlere (mediane) Zeiten bis zum Erreichen der Kontinenz werden durch ein proportional-hazards-model geschätzt.

Erreichen von Kontinenz und Tod sind mathematisch gesehen konkurrierende Ereignisse. D. h. für einen Patienten, welcher verstorben ist ohne Kontinenz erreicht zu haben, gilt die Zeit bis zum Tod hinsichtlich Kontinenz als "zensiert". Dies wird einerseits aber selten vorkommen. Andererseits ist fast auszuschließen, dass hierbei zwischen beiden Armen eine große Schieflage besteht. Methoden der "competing risks analysis" sind deshalb verzichtbar.

Zu den Zeitpunkten 1, 3, 6 und 12 Monate werden Raten (binäre Merkmale) zwischen den Behandlungsgruppen mit dem  $\chi^2$ -Test verglichen, bei geringen Häufigkeiten mit Fisher's exact test. Kontinuierliche Größen werden mit dem Mann-Whitney U-Test für zwei bzw. dem H-Test nach Kruskal-Wallis für mehr als 2 Gruppen verglichen. Dabei werden die Fragebogenskalen als quasi-kontinuierlich betrachtet. Für die Behandlungseffekte werden Konfidenzintervalle berechnet.

Die Analyse der Längsschnittdaten erfolgt durch ANOVA mit wiederholten Messungen. Posthoc-Tests sichern dabei das Fehlerniveau beim multiplen Testen. Ebenso mit verallgemeinerten bzw. allgemeinen linearen Modellen wird die Assoziation verschiedener Risikofaktoren (BMI, nerverhaltende OP usw.) mit den Endpunkten untersucht. Dabei soll auch der Einfluss des Operateurs bzw. seiner Erfahrung als Kofaktor in multivariaten Modellen getestet werden. Verschwindet ein evtl. vorher vorhandener Behandlungseffekt nach Adjustierung auf die Operateure (bzw. ihre Erfahrung), so lässt sich schließen, dass nicht die Roboter-Assistenz, sondern eher die Übung des Operateurs den Unterschied in der Kontinenz bewirkt hat.

Es ist vorgesehen, die Untergruppen hinsichtlich nerverhaltender Operation (vgl. A1, A2, A3 in 9.1) zumindest deskriptiv auszuwerten. Die Ersetzung fehlender Werte ist nur in Ausnahmefällen vorgesehen. Details hierzu werden in einem Statistischen Analyseplan vor Studienende festgelegt.

#### 9.5.2 Auswertbarkeit eines Patienten

Als auswertbar gilt jeder randomisierte Patient, welcher mit LRPE bzw. R-LRPE operiert wurde. Im Detail entscheidet das Vorhandensein bestimmter Werte, ob der Patient in spezielle Analysen einbezogen werden kann oder nicht (s. 9.5.1).

# 9.6 Zwischenauswertungen

Um bei Überlegenheit ein vorzeitiges Studienende zu ermöglichen, wird eine Zwischenauswertung des primären Endpunkts vorgesehen, wenn die Hälfte der geplanten Patienten ihr 3-Monats-Follow-up abgeschlossen hat. Nach Plan wäre das am Ende von 21 Monaten. Nach 39 Monaten (3 Jahre Rekrutierung und 3 Monate Follow-up) wird der Termin für den primären Endpunkt erreicht. Tabelle 6 gibt die beim Test verwendeten Abbruchgrenzen nach Kim/deMets für beide Zeitpunkte sowie Fehler 1. Art und Power an.

| Tabelle 6 | Abbrucngrenzen |
|-----------|----------------|

| | Abbruch | grenzen | Kumulativ | |
|-----------|---------|---------|-----------|-------|
| | untere | obere | Alpha | Power |
| 21 Monate | -2.44 | 2.44 | 0.014 | 0.360 |
| 39 Monate | -2.03 | 2.03 | 0.050 | 0.800 |

D. h., angenommen es liege tatsächlich ein Unterschied der 3-Monats-Kontinenzraten von 44% vs. 34% vor, besteht eine Wahrscheinlichkeit von 36%, dass die Studie vorzeitig beendet werden kann. Ein vorzeitiger Abbruch der Studie wegen Futility ist nicht vorgesehen.

#### 9.7 Endauswertung

Die Endauswertung der Daten bis zum 12 Monats-Follow-up erfolgt, nachdem der letzte Patient die 12 Monats-Visite beendet hat und alle Queries beantwortet sind. Die Auswertung der onkologischen Daten (24 und 36 Monate postoperativ) erfolgt, nachdem die entsprechenden Daten für den letzten Patienten eingeholt und überprüft wurden und die Datenbank für diesen Datenbereich geschlossen worden ist. Die Datenerhebung für das 36 Monats-Follow-up wird abgeschlossen, wenn für alle Patienten das 24-Monats-Follow-up beendet ist, d. h. nach 5 Jahren Datenerhebung. Zu diesem Zeitpunkt haben 2/3 der Patienten das 36-Monats-Follow-up erreicht.

Die Verfahren zur Auswertung werden detailliert vor Studienende in einem Statistischen Analyseplan festgelegt.

# 10 Datenmanagement

### 10.1 Prüfbögen (Case Report Forms - CRF)

Für jeden Patienten wird durch die Studienzentrale ein papierbasierter CRF erstellt, in den die anonymisierten Befunde aller Untersuchungen der jeweiligen Visite eingetragen werden. Die entsprechenden Originalbefunde finden Eingang in die Patientenakte (stationär).

Der CRF wird auf "non-copy carbon Paper" gedruckt, so dass der Originalbogen zur Dateneingabe an die Studienzentrale in Leipzig gesendet werden kann. Die Kopie verbleibt im Prüfarztordner im Prüfzentrum. Die Versendung aller Follow-Up Bögen sowie die komplette Dateneingabe erfolgen durch die Studienzentrale.

Die Bögen zur Dokumentation unerwünschter und schwerwiegender unerwünschter Ereignisse erstellt die Studienzentrale zusammen mit dem ZKS Leipzig - KKS.

Alle Einträge im CRF werden deutlich lesbar mit dunklem Kugelschreiber vorgenommen, um die Lesbarkeit von Durchschlägen oder Kopien zu gewährleisten. Korrekturen werden so durchgeführt, dass der Originaleintrag lesbar bleibt und mit Datum und Initialen der zur Korrektur berechtigten Person abgezeichnet wird. Sollten Daten oder Einträge fehlen, so muss dieses begründet werden. Alle relevanten CRF-Seiten werden durch den Hauptprüfer oder einen Prüfer auf Vollständigkeit und Korrektheit kontrolliert und abgezeichnet. Die Unterschrift dient der Verifizierung der CRF-Einträge.

Als Quelldaten (source data) im Sinne der ICH-Richtlinie E6 werden alle Daten der Patientenakte, sowie routinemäßig erhobene Daten und Laborberichte der einzelnen Untersuchungen betrachtet.

Die Originale der CRF-Seiten werden nach jeweils fünf aus dem Krankenhaus entlassenen Patienten zur Dateneingabe an die Studienzentrale gesendet. Die Durchschläge verbleiben im Prüfarztordner im Prüfzentrum.

## 10.2 Datenmanagement

Das Datenmanagement erfolgt unter Verwendung des Studienmanagement-Tools eResearchNetwork. Für die Erstellung der Studiendatenbank wird vom verantwortlichen Projektmanager in Zusammenarbeit mit dem Biometriker ein Pflichtenheft formuliert, das dem Datenbankprogrammierer als Basis für die Erstellung der Datenbankanwendung dient. Vor Freigabe wird die Datenbankanwendung auf Fehler getestet und validiert, der Vorgang der Validierung wird schriftlich dokumentiert.

Die auf den CRFs erfassten Daten werden über Eingabemasken in der eResearch-Datenbank in der Studienzentrale erfasst. Die eingegebenen Daten werden täglich über vorprogrammierte, automatische Checks auf Vollständigkeit, Konsistenz und Plausibilität überprüft. Rückfragen (Queries) werden zeitnah in schriftlicher Form an die Prüfzentren bzw. die verantwortlichen Monitore übermittelt.

Es erfolgt eine tägliche Komplettsicherung aller Daten. Durch den Einsatz eines hierarchischen auf Rollen basierenden Zugriffskonzeptes ist ein unberechtigter Zugriff auf die Patientendaten unmöglich. Die Anonymität der Daten im Rahmen von Auswertungen ist sichergestellt. Jede Änderung an den Daten, z.B. aufgrund der Einarbeitung von beantworteten Rückfragen, wird über einen automatischen Audittrail in der Datenbank dokumentiert.

Am Studienende wird nach Eingabe aller Eintragungen die Datenbank geschlossen. Dieser Vorgang wird von der Studienzentrale dokumentiert. Für die Auswertungen wird die Software IBM SPSS Statistics (Version 20) verwendet.

Die im Rahmen der Studie erhobenen Patientendaten werden in pseudonymisierter Form mit Hilfe einer Identifikations-Nummer elektronisch gespeichert und ausgewertet. Die Studiendaten sind vor fremden Zugriff geschützt; nur Mitarbeiter der Studie dürfen auf diese zugreifen. Diese Mitarbeiter sind zur Verschwiegenheit verpflichtet. Der Hauptprüfer des Zentrums führt eine Patientenidentifikationsliste, in der die Patientenidentifikationsnummern mit dem vollen Patientennamen verbunden sind. Diese Liste ist absolut vertraulich zu behandeln und darf das Prüfzentrum nicht verlassen. Die Patientenidentifikationsliste ist nach Studienende mindestens zehn Jahre zu archivieren.

# 10.3 Archivierung

Alle relevanten Studienunterlagen (Trial Master File), die elektronisch erfassten Daten, die Originale aller CRFs, Zwischen- und Abschlussbericht werden mindestens 10 Jahre nach Abschluss der Studie in der Studienzentrale, Klinik und Poliklinik für Urologie in Leipzig, aufbewahrt.

In den Prüfzentren werden der Prüfarztordner, die Patientenidentifikationsliste, die unterschriebenen Einwilligungserklärungen, Kopien aller CRFs und die Patientenakten mindestens 10 Jahre nach Abschluss der Studie aufbewahrt. Verlangen hausinterne Regelungen oder andere Gesetzgebungen eine längere Aufbewahrungsfrist, ist diese zu berücksichtigen.

# 11 Qualitätssicherung

# 11.1 Zugang zu Quelldaten

Aufgrund gesetzlicher Regelungen zur Sicherung der Datenqualität und zur Überwachung der Studiendurchführung am Zentrum sind die Prüfärzte verpflichtet, autorisierten Dritten Einsicht in die Patientenakten (Quelldaten) zu gewährleisten. Dazu zählen Monitore, Auditoren und weitere Beauftragte des Auftraggebers, Mitarbeiter der zuständigen Überwachungsbehörde oder der Bundesoberbehörde. Diese Personen sind zur Verschwiegenheit verpflichtet.

# 11.2 Monitoring

Zur Überwachung der Prüfzentren wird im Verlauf der Studie ein on-site Monitoring durch Mitarbeiter des KKS Leipzig durchgeführt.

Im Rahmen dieser Monitoring-Besuche werden alle studienrelevanten Dokumente kontrolliert und ggf. aktualisiert und es wird ein 100%tiger Quelldatenvergleich der Eckdaten (z. B. Patientenexistenz, Vorliegen der Einverständniserklärung) zur Überprüfung der Einverständniserklärungen sowie ein partieller Quelldatenvergleich der weiteren Einträge in den CRFs der Studienteilnehmer durchgeführt.

Zum Studienabschluss sind Abschlussbesuche in allen Prüfzentren geplant.

Zur Durchführung des Monitorings ermöglichen die Prüfer den Zutritt zu den Räumlichkeiten der Studiendurchführung und Zugriff auf die Akten aller Studienteilnehmer zur Gewährleistung eines vollständigen Quelldatenvergleichs.

Die exakte Planung und Durchführung des Monitorings basiert auf den dafür verfügbaren SOPs des KKS Leipzig und wird in einem noch zu erstellenden Monitoringmanual genauer beschrieben.

# 12 Ethische und regulatorische Grundlagen

#### 12.1 GCP-Erklärung

Die Studie wird nach dem aktuellen Stand der medizinisch-wissenschaftlichen Erkenntnisse durchgeführt und alle an der Studie Beteiligten (Auftraggeber, Bevollmächtigte und Auftragnehmer des Auftraggebers, Prüfer etc.) verpflichten sich, die klinische Prüfung nach den

Vorgaben der nationalen Gesetze, den Anforderungen der ICH Guideline for Good Clinical Practice (GCP) E6 vom Juni 1996 und der CPMP/ICH/135/95 vom September 1997 durchzuführen und die Empfehlungen der aktuellen Deklaration von Helsinki (Version Fortaleza, Brasilien, Oktober 2013) zu beachten.

### 12.2 Antragstellung

Gemäß den Vorgaben der Musterberufsordnung der Ärzte §15 wird die klinische Prüfung vor Beginn den zuständigen Ethikkommissionen der teilnehmenden Prüfärzte zur Beratung vorgelegt. Hierzu wird das bereits vorhandene primäre EK-Votum des Studienleiters den Antragsunterlagen beigelegt.

# 13 Gesetzliche und administrative Regelungen

# 13.1 Studiendurchführung nach Prüfplan

Die hier dargestellte klinische Prüfung wird entsprechend den Anforderungen von ICH-GCP und den geltenden gesetzlichen Bestimmungen (MPG) geplant, durchgeführt und ausgewertet.

Protokollverletzungen sind sämtliche Abweichungen von den Anweisungen und Abläufen, die in diesem Prüfplan beschrieben werden. Dazu gehören:

- fehlende Untersuchungen bzw. Durchführung dieser zum falschen Zeitpunkt
- fehlende Compliance
- Behandlung nicht entsprechend dem Randomisationsergebnis
- Nutzung unerlaubter Medizinprodukte

Nachdem ein Studienteilnehmer in die Studie aufgenommen wurde, liegt es in der Verantwortung des Prüfers Protokollverletzungen zu vermeiden, um den Patienten in der Studie zu halten.

Schwerwiegende Protokollverletzungen werden unverzüglich an die Studienleitung gemeldet. Die Einschätzung von Protokollverletzungen erfolgt im Monitoring Manual. Alle Protokollverletzungen werden dokumentiert und vor der statistischen Auswertung der Studie mit dem verantwortlichen Biometriker diskutiert.

Der Prüfer muss sicherstellen, dass alle erhobenen Daten entsprechend dem Prüfplan dokumentiert werden. Kleinere Abweichungen sind im Arbeitsalltag sicherlich nicht zu vermeiden, müssen allerdings mit einer Begründung dokumentiert werden.

### 13.2 Nachträgliche Prüfplanänderungen

Jede nachträgliche Prüfplanänderung (Protokoll-Amendments, technische Änderungen) darf nur durch die Studienleitung vorgenommen werden (ggfs. in Absprache mit der Biometrie) und muss im Trial Master File mit Datum vermerkt und allen Studienbeteiligten schriftlich mitgeteilt werden.

Protokoll-Amendments: Eingreifende Änderungen von Studiendesign, Studienablauf oder Auswertungsverfahren sind als Prüfplanamendment bei der federführenden Ethikkommission einzureichen. Eine ggf. erforderliche Anpassung von Dokumenten (z.B. Patienteninformation, Dokumentationsbögen) erfolgt durch die Studienleitung.

Technische Änderungen des Protokolls: Änderungen, die aus organisatorischen oder administrativen Gründen erforderlich sind, bedürfen keiner Einreichung bei der Ethikkommission. Dazu gehört auch die Korrektur nachträglich festgestellter formaler Fehler des Protokolls.

## 13.3 Verantwortlichkeit der Prüfer und Prüferverträge für klinische Studien

Die Prüferverträge für klinische Studien müssen in jedem Studienzentrum vom Hauptprüfer unterschieben werden und sind vor Beginn der Studientätigkeit des Zentrums an die Studienzentrale zurückzuschicken.

Der Hauptprüfer jedes Zentrums ist für die Weiterleitung der CRFs, Todesmeldungen, meldepflichtigen unerwünschten Ereignisse und Abweichungen vom Studienprotokoll an die Studienzentrale verantwortlich. Alle Studiendokumente (z.B. Studienprotokoll, Bescheid der federführenden Ethikkommission des Leiters der Klinischen Prüfung) müssen der lokalen Ethikkommission der Prüfzentren gemäß den örtlichen Vorschriften unverzüglich eingereicht werden. Kopien aller wichtigen Unterlagen über etwaige Maßnahmen seitens der lokalen Ethikkommission in Bezug auf diese klinische Studie müssen an die Studienzentrale weitergeleitet werden. Alle Berichte und Dokumente unterliegen den Anforderungen zur Dokumentenaufbewahrung.

### 13.4 Finanzierung und Versicherungen

Die Förderung der Studie wird bei der deutschen Krebshilfe beantragt.

Es wird keine Probandenversicherung benötigt, da es sich hierbei um eine klinische Prüfung nach §23b MPG handelt, die Studie im Rahmen der Zweckbestimmung der bereits bestehenden CE-Kennzeichnung und ohne zusätzliche invasive oder belastende Untersuchungen für die Patienten durchgeführt wird, und hier die Produkthaftpflicht des Medizinproduktes greift. Die endgültige Bewertung erfolgt durch die zuständige Ethikkommission.

#### 13.5 Publikationsvereinbarungen und Registrierung

Die Studie wird bei "Controlled Clinical Trials" (www.clinicaltrials.gov) angemeldet.

Die finale Publikation der Studienergebnisse erfolgt durch die Studienzentrale auf der Grundlage der durchgeführten statistischen Analysen. Alle teilnehmenden Zentren werden bei Veröffentlichungen beteiligt. Ein Entwurfsmanuskript wird an das ZKS Leipzig - KKS und an alle Koautoren zur Prüfung gegeben. Nach der Überprüfung durch den Biometriker und die anderen Koautoren wird das Manuskript bei wissenschaftlichen Zeitschriften mit peer review zur Veröffentlichung eingereicht. Die Veröffentlichung der Studienergebnisse erfolgt unabhängig davon, wie die Ergebnisse ausfallen.

Die Erstautorenschaft wird durch den klinischen Studienleiter und/oder den Projektmanager gestellt. Der Hauptprüfer der anderen Zentren, der Biometriker, wissenschaftlich aktiv beitragende Personen und Prüfer, die mehr als 5% der auswertbaren Patienten eingebracht haben, werden als Koautoren benannt. Die Reihenfolge der Autorenschaft richtet sich nach der aktiven Teilnahme an der Durchführung der Studie und der Anzahl der eingebrachten Studienpatienten. Die Seniorautorenschaft liegt bei der Klinik mit der höchsten eingebrachten Zahl an auswertbaren Patienten.

Jegliche Veröffentlichungen, Abstracts und Präsentationen, die auf eingeschlossenen Studienpatienten basieren, müssen von der Studienleitung genehmigt werden. Dies gilt für jeden registrierten/randomisierten Studienpatienten oder jede Subgruppe von Studienpatienten. Teilergebnisse bzw. Auswertungen von Forschungsfragen, denen die Daten einzelner Kliniken zugrunde liegen, sind mit Genehmigung durch die Studienleitung Leipzig möglich.

Erstautorschaft kann dann von der jeweiligen Klinik gestellt werden. Eine solche Veröffentlichung kann weder den Vergleich zwischen den randomisierten Behandlungsgruppen (LRPE vs. R-LRPE) noch eine Analyse der Endpunkte der Studie umfassen, solange keine endgültigen Ergebnisse der Studie veröffentlicht wurden.

Vorab veröffentlichte Publikationen oder Präsentationen der Studie können demographische Daten, Gesamtergebnisse oder prognostische Analysen enthalten, jedoch keine Vergleiche zwischen den beiden randomisierten Therapiearmen, bevor die Rekrutierung nicht abgeschlossen ist.

Im Falle der Veröffentlichung von Projektergebnissen, Projektmitteilungen, Tagungsbeiträgen und Präsentationen wird auf die finanzielle Förderung durch die DKH hingewiesen.

# 14 Literatur

- Aaronson NK, Ahmedzai S, Bergman B, Bullinger M, Cull A, Duez NJ, Filiberti A, Flechtner H, Fleishman SB, de Haes JC. The European Organization for Research and Treatment of Cancer QLQ-C30: a quality-of-life instrument for use in international clinical trials in oncology. J Natl Cancer Inst 1993; 85 (5): 365-376.
- Agarwal PS, Sammona J, Bhandari A, Dabaja A, Diaz M, Dusik-Fenton S, Satyanarayana R, Simone A, Trinh Q, Baize B, Menon M. Safety profile of robot-assisted radical prostatectomy: a standardized report of complications in 3317 patients. Eur Urol 2011; 59: 684-698.
- Asimakopoulos AD, Pereira Fraga CT, Annino FP, Patrizio C, Calado AA, Mugnier C: Randomized Comparison between Laparoscopic and Robot-Assisted Nerve-Sparing Radical Prostatectomy. J Sex Med 2011; 8 (5): 1503–1512.
- Badani KK, Kaul S, Menon M: Evolution of robotic radical prostatectomy: assessment after 2766 procedures. Cancer 2007; 110 (9):1951-8.
- Berryhill R, Jhaveri J, Yadav R, Leung R, Rao S, El-Hakim A, Tewari A. Robotic Prostatectomy: A Review of Outcomes Compared with Laparoscopic and Open Approaches. Urology 2008; 72 (1): 15–23.
- Börgermann C, Kaufmann A, Sperling H, Stöhrer M, Rübben H. Therapie der Belastungsinkontinenz beim Mann. Dtsch Arztebl Int 2010; 107 (27): 484–491.
- Clavien PA, Barkun J, de Oliveira ML, Vauthey JN, Dindo D, Schulick RD, de Santibanes E, Pekolj J, Slankamenac K, Bassi C, Graf R, Vonlanthen R, Padbury R, Cameron JL, Makuuchi M. The Clavien-Dindo Classification of Surgical Complications Five-Year Experience. Annals of Surgery 2009; 250 (2): 187-196.
- Dindo D, Demartines N, Clavien PA. Classification of surgical complications A new proposal with evaluation in a cohort of 6336 patients and results of a survey. Annals of Surgery 2004; 240 (2): 205-213.
- Do HM, Holze S, Qazi H, Dietel A, Häfner T, Liatsikos E, Stolzenburg J-U (2012): Radikale Prostatektomie. Pro laparoskopisch. Der Urologe, 51(5): 617-623. Fayers P, Aaronson NK, Bjordal K. *EORTC QLQ-C30 Scoring Manual*. Brussels, EORTC Study Group on Quality of Life. 1995.
- Ficarra V, Novara G, Artibani W, Cestari A, Galfano A, Graefen M, Guazzoni G, Guillonneau B, Menon M, Montorsi F, Patel V, Rassweiler J, Van Poppel H. Retropubic, laparoscopic, and robot-assisted radical prostatectomy: a systematic review and cumulative analysis of comparative studies. Eur Urol 2009; 55 (5): 1037-1063.
- Fleiss JL, Levin B, Paik MC. Statistical Methods for Rates and Proportions. Third Edition. John Wiley & Sons. New York 2003.
- Guillonneau B, Vallancien G: Laparoscopic radical prostatectomy: the Montsouris experience. J Urol 2000; 163 (2): 418–422.
- Hakenberg O. Ein Leben ohne Roboter. Was bleibt dem Urologen? Urologe 2010; 49 (8): 922-924.
- Hakimi A, Blitstein J, Feder M, Shapiro E, Ghavamian R. Direct Comparison of Surgical and Functional Outcomes of Robotic-Assisted Versus Pure Laparoscopic Radical Prostatec-

- tomy: Single-Surgeon Experience. Urology. 2009; 73 (1): 119-23.
- Hakimi A, Faleck DM, Sobey S, Ioffe E, Rabbani F, Donat SM, Ghavamian R. Assessment of complication and functional outcome reporting in the minimally invasive prostatectomy literature from 2006 to the present. BJU International 2011; 109: 26-30.
- Heidenreich A, Aus G, Abbou CC, Bolla M, Joniau S, Matveev V, Schmid HP, Zattoni F, European Association of Urology (EAU). EAU guidelines on prostate cancer. Arnhem: EAU; 2007.
- Hermann C, Buss U, Snaith RP. HADS-D: Hospital Anxiety and Depression Scale Deutsche Version. Ein Fragebogen zur Erfassung von Angst und Depressivität in der somatischen Medizin. Bern, 1995.
- Herrmann TR, Rabenalt R, Stolzenburg JU, Liatsikos EN, Imkamp F, Tezval H, et al. Oncological and functional results of open, robot-assisted and laparoscopic radical prostatectomy: does surgical approach and surgical experience matter? World J Urol 2007; 25: 149-160.
- Holze S, Koehler N, Gansera L, Rebmann U, Truss MC, Roth S, Scholz H-J, Fahlenkamp D, Thiel R, Casey RG, Braehler E, Stolzenburg J-U. Quality of life after retropubic and endoscopic extraperitoneal radical prostatectomy: A prospective multicentre study. J Psychosoc Onc (eingereicht) 2011.
- Jennison C, Turnbull BW. Group Sequential Methods with Applications to Clinical Trials.Boca Raton: Chapman and Hall, 2000.
- Kang DC, Hardee MJ, Fesperman SF, Stoffs TL, Dahma P. Low Quality of Evidence for Robot-Assisted Laparoscopic Prostatectomy: Results of a Systematic Review of the Published Literature. Eur Urol 2010; 57: 930-937.
- King M. The interpretation of scores from the EORTC quality of life questionnaire QLQ-C30. Quality of Life Research, 1995; 5(6), 555-567.
- Kirby R, Montorsi F, Gontero P, Smith JA. Radical prostatectomy: From open to robotic. Informa Healthcare, London, 2007.
- Köhler N, Gansera L, Stolzenburg JU, Rebmann U, Truss MC, Roth S, Scholz HJ, Fahlenkamp D, Thiel R, Liatsikos E, Braehler E, Holze S: Early continence in patients with localized prostate cancer. A comparison between open retropubic (RRPE) and endoscopic extraperitoneal radical prostatectomy (EERPE). Urologic Oncology, 2011 (im Druck).
- Krambeck AE, DiMarco DS, Rangel LJ. Radical prostatectomy for prostatic adenocarcinoma: a matched comparison of open retropubic and robot-assisted techniques. BJU Int. 2009; 103 (4): 448-53.
- Link RE, Su LM, Sullivan W, Bhayani, SB, Pavlovich, CP. Link Health related quality of life before and after laparoscopic radical prostatectomy. J Urol 2005; 173 (1): 175-179.
- Machin D, Campbell M, Fayers P, Pinol A: Sample Size Tables for Clinical Studies. Blackwell Science, Oxford, 1997.
- Mulhall JP, Goldstein I, Bushmakin AG, Cappelleri J, Hvidsten K. Validation of the erection hardness score. J Sex Med 2009; 4 (6): 1626-1634.
- Murphy DG, Kerger M, Crowe H. Operative details and oncological and functional outcome of robotic-assisted laparoscopic radical prostatectomy: 400 cases with a minimum of 12

- months follow-up. Eur Urol 2009; 55 (6): 1358-66.
- Murphy DG, Bjartell A, Fivarra V, Graefen M, Haese A, Montironi R, Montorsi F, Moul, J, Novara G, Sauter G, Sulser T, van der Poel H. Downsides of Robot-assisted Laparoskopic Radical Prostatectomy: Limitations and Complications. Eur Urol 2010; 57: 735-746.
- Osoba D, Rodrigues G, Myles J, Zee B, Pater J. Interpreting the significance of changes in health-related quality-of-life scores. Journal of Clinical Oncology 1998; 16 (1), 139-144.
- Patel VR, Coelho RF, Chauhan S. Continence, potency and oncological outcomes after robotic-assisted radical prostatectomy: early trifecta results of a high-volume surgeon. BJU Int 2010; 106 (5): 696-702.
- Pietrow PK, Parekh DJ, Smith JA, Shyr Y, Cookson M S. Health related quality of life assessment after radical prostatectomy in men with prostate specific antigen only recurrence. Journal of Urology 2011; 166 (6): 2286-2290.
- Pockock SJ, Simon R. Sequential treatment assignment with balancing for prognostic factors in the controlled clinical trial. Biometrics 1975; 31 (1): 103-115.
- Rassweiler J, Stolzenburg J, Sulser T. Laparoscopic radical prostatectomy--the experience of the German Laparoscopic Working Group. Eur Urol 2006; 49 (1): 113-9.
- Robert-Koch-Institut. Krebs in Deutschland 2005/2006. Häufigkeiten und Trends. Robert-Koch-Institut, Berlin, 2010.
- Rodrigues G, Bezjak A, Osoba D, Catton P, Tsuji D, Taylor D, Warde P. The relationship of changes in EORTC QLQ-C30 scores to ratings on the Subjective Significance Questionnaire in men with localized prostate cancer. Quality of Life Research, 2004; 13 (7): 1235-1246.
- Rosen RC, Cappelleri JC, Smith MD, Lipsky J, Peña BM. Development and evaluation of an abridged 5 version of the International Index of Erectile Function (IIEF-5) as a diagnostic tool for erectile dysfunction. Int J Impot Res 1999; 11: 319–26.
- S3 Leitlinie Interdisziplinäre Leitlinie der Qualität S3 zur Früherkennung, Diagnose und Therapie der verschiedenen Stadien des Prostatakarzinoms. Deutsche Gesellschaft für Urologie e. V. 2011.
- Stolzenburg JU, Rabenalt R, Do M, Lee B, Truss MC, Schwaibold H, Burchardt M, Jonas U, Liatsikos EN. Categorisation of complications of endoscopic extraperitoneal and laparoscopic transperitoneal radical prostatectomy. World J Urol 2006; 24 (1): 88-93.
- Stolzenburg J-U, Türk IA, Liatsikos E. Laparoscopic and Robot-Assisted Surgery in Urology. Atlas of Standard Procedures. Berlin: Springer 2011.
- Twiss CO, Fischer MC, Nitti VW. Comparison between reduction in 24-hour pad weight, International Consultation on Incontinence-Short Form (ICIQ-SF) score, International Prostate Symptom Score (IPSS), and post-operative Patient Global Impression of Improvement (PGI-I) score in patient evaluation after male perineal sling. Neurourol Urodyn 2007; 26 (1): 8-13.
- Van Andel G, Bottomley A, Fossa SD, Efficace F, Coens C, Guerif S, Kynaston H, Gontero P, Thalmann G, Akdas A, D'Haese S, Aaronson NK. An international field study of the EORTC QLQ-PR25: A questionnaire for assessing the health-related quality of life of patients with prostate cancer. Eur J Cancer 2008; 44 (16): 2418-2424.

- Wiltink J, Hauck EW, Phadayanon M, Weidner W, Beutel ME. Validation of the German version of the International Index of Erectile Function (IIEF) in patients with erectile dysfunction, Peyronie's disease and controls. Int J Impot Res 2003; 15 (3): 192-197.
- Zahiri CA, Schmalzried TP, Szuszczewicz ES, Amstutz HC. Assessing activity in joint replacement patients. J Arthroplasty. 1998;13:890–895.